CLINICAL TRIAL: NCT01131676
Title: A Phase III, Multicentre, International, Randomised, Parallel Group, Double Blind Cardiovascular Safety Study of BI 10773 (10 mg and 25 mg Administered Orally Once Daily) Compared to Usual Care in Type 2 Diabetes Mellitus Patients With Increased Cardiovascular Risk
Brief Title: BI 10773 (Empagliflozin) Cardiovascular Outcome Event Trial in Type 2 Diabetes Mellitus Patients (EMPA-REG OUTCOME).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.25; 2009-016178-33 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

ARMS (3):
- BI 10773 low dose (Experimental): BI 10773 tablets once daily
  Interventions: Drug: BI 10773 low dose; Drug: Placebo BI 10773 high dose
- BI 10773 high dose (Experimental): BI 10773 tablets once daily
  Interventions: Drug: BI 10773 high dose; Drug: Placebo BI 10773 low dose
- Placebo (Placebo Comparator): Placebo tablets matching BI 10773
  Interventions: Drug: Placebo BI 10773 high dose; Drug: Placebo BI 10773 low dose

INTERVENTIONS:
Drug: BI 10773 low dose — BI 10773 tablets once daily
  Arms: BI 10773 low dose
Drug: Placebo BI 10773 high dose — Placebo tablets identical to BI 10773
  Arms: Placebo
Drug: BI 10773 high dose — BI 10773 tablets once daily
  Arms: BI 10773 high dose
Drug: Placebo BI 10773 low dose — Placebo tablets identical to BI 10773
  Arms: BI 10773 high dose
Drug: Placebo BI 10773 low dose — Placebo tablets identical to BI 10773
  Arms: Placebo
Drug: Placebo BI 10773 high dose — Placebo tablets identical to BI 10773
  Arms: BI 10773 low dose

SUMMARY:
The aim of the present study is to investigate the safety of BI 10773 treatment in patients with Type 2 Diabetes Mellitus and high cardiovascular risk.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of type 2 diabetes mellitus prior to informed consent
2. Male or female patients on diet and exercise regimen who are drug naive or pre treated with any background therapy. Antidiabetic therapy has to be unchanged for 12 weeks prior to randomization.
3. Glycosylated haemoglobin (HbA1c) of >= 7.0% and <=10% for patients on background therapy or HbA1c >= 7.0% and <= 9.0% for drug naive patients
4. Age >= 18 years
5. Body Mass index <= 45 at Visit 1
6. Signed and dated informed consent
7. High cardiovascular risk

Exclusion criteria:

1. Uncontrolled hyperglycaemia with a glucose level >240 mg/dl (>13.3 mmol/L) after an overnight fast during placebo run-in and confirmed by a second measurement (not on the same day)
2. Indication of liver disease, defined by serum levels of either alanine aminotransferase (ALT), aspartate aminotransferase ALT or alkaline phosphatase above 3 x upper limit of normal (ULN) as determined at screening and/or run in.
3. Planned cardiac surgery or angioplasty within 3 months
4. Impaired renal function, defined as Glomerular Filtration Rate <30 ml/min (severe renal impairment, Modification of Diet in Renal Disease formula) during screening or run in.
5. Bariatric surgery within the past two years and other gastrointestinal surgeries that induce chronic malabsorption
6. Blood dyscrasias or any disorders causing haemolysis or unstable Red Blood Cell (e.g. malaria, babesiosis, haemolytic anemia)
7. Medical history of cancer (except for basal cell carcinoma) and/or treatment for cancer within the last 5 years
8. Contraindications to background therapy according to the local label
9. Treatment with anti-obesity drugs (e.g. sibutramine, orlistat) 3 months prior to informed consent or any other treatment at the time of screening (i.e. surgery, aggressive diet regimen, etc.) leading to unstable body weight
10. Current treatment with systemic steroids at time of informed consent or change in dosage of thyroid hormones within 6 weeks prior to informed consent or any other uncontrolled endocrine disorder except type 2 diabetes mellitus
11. Pre-menopausal women (last menstruation <+ 1 year prior to informed consent) who:

    * are nursing or pregnant or
    * are of child-bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the study and do not agree to submit to periodic pregnancy testing during participation in the trial. Acceptable methods of birth control include tubal ligation, transdermal patch, intra uterine devices/systems, oral, implantable or injectable contraceptives, sexual abstinence, double barrier method and vasectomised partner
12. Alcohol or drug abuse within the 3 months prior to informed consent that would interfere with trial participation or any ongoing condition leading to a decreased compliance to study procedures or study drug intake
13. Participation in another trial with an investigational drug within 30 days prior to informed consent
14. Any other clinical condition that would jeopardize patients safety while participating in this clinical trial
15. Acute coronary syndrome, stroke or TIA within 2 months prior to informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7064 (Actual)
Dates: Start 2010-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (615):
- United States (170):
  - 1245.25.10043 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1245.25.10121 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1245.25.10037 Boehringer Ingelheim Investigational Site, Huntsville, Alabama
  - 1245.25.10124 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 1245.25.10015 Boehringer Ingelheim Investigational Site, Little Rock, Alaska
  - 1245.25.10056 Boehringer Ingelheim Investigational Site, Gilbert, Arizona
  - 1245.25.10175 Boehringer Ingelheim Investigational Site, Peoria, Arizona
  - 1245.25.10072 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 1245.25.10048 Boehringer Ingelheim Investigational Site, Harrisburg, Arkansas
  - 1245.25.10035 Boehringer Ingelheim Investigational Site, Anaheim, California
  - 1245.25.10103 Boehringer Ingelheim Investigational Site, Encino, California
  - 1245.25.10158 Boehringer Ingelheim Investigational Site, Fresno, California
  - 1245.25.10126 Boehringer Ingelheim Investigational Site, Harbor City, California
  - 1245.25.10058 Boehringer Ingelheim Investigational Site, Huntington Park, California
  - 1245.25.10001 Boehringer Ingelheim Investigational Site, Lancaster, California
  - 1245.25.10102 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1245.25.10047 Boehringer Ingelheim Investigational Site, Los Gatos, California
  - 1245.25.10118 Boehringer Ingelheim Investigational Site, Palm Springs, California
  - 1245.25.10061 Boehringer Ingelheim Investigational Site, Riverside, California
  - 1245.25.10040 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1245.25.10055 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1245.25.10193 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1245.25.10027 Boehringer Ingelheim Investigational Site, Santa Rosa, California
  - 1245.25.10074 Boehringer Ingelheim Investigational Site, Stockton, California
  - 1245.25.10083 Boehringer Ingelheim Investigational Site, Valencia, California
  - 1245.25.10144 Boehringer Ingelheim Investigational Site, Colorado Springs, Colorado
  - 1245.25.10085 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1245.25.10153 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1245.25.10066 Boehringer Ingelheim Investigational Site, Norwalk, Connecticut
  - 1245.25.10038 Boehringer Ingelheim Investigational Site, Waterbury, Connecticut
  - 1245.25.10068 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 1245.25.10094 Boehringer Ingelheim Investigational Site, Bradenton, Florida
  - 1245.25.10190 Boehringer Ingelheim Investigational Site, Brooksville, Florida
  - 1245.25.10209 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1245.25.10212 Boehringer Ingelheim Investigational Site, Cooper City, Florida
  - 1245.25.10200 Boehringer Ingelheim Investigational Site, Delray Beach, Florida
  - 1245.25.10033 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1245.25.10202 Boehringer Ingelheim Investigational Site, Hallandale, Florida
  - 1245.25.10062 Boehringer Ingelheim Investigational Site, Hialeah, Florida
  - 1245.25.10063 Boehringer Ingelheim Investigational Site, Hialeah, Florida
  - 1245.25.10157 Boehringer Ingelheim Investigational Site, Hialeah, Florida
  - 1245.25.10089 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1245.25.10019 Boehringer Ingelheim Investigational Site, Longwood, Florida
  - 1245.25.10168 Boehringer Ingelheim Investigational Site, Maitland, Florida
  - 1245.25.10018 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1245.25.10039 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1245.25.10184 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1245.25.10123 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1245.25.10201 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1245.25.10025 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 1245.25.10042 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 1245.25.10147 Boehringer Ingelheim Investigational Site, Port Charlotte, Florida
  - 1245.25.10198 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 1245.25.10203 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 1245.25.10104 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1245.25.10178 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1245.25.10211 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1245.25.10023 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 1245.25.10174 Boehringer Ingelheim Investigational Site, Columbus, Georgia
  - 1245.25.10141 Boehringer Ingelheim Investigational Site, Riverdale, Georgia
  - 1245.25.10067 Boehringer Ingelheim Investigational Site, Roswell, Georgia
  - 1245.25.10022 Boehringer Ingelheim Investigational Site, Honolulu, Hawaii
  - 1245.25.10092 Boehringer Ingelheim Investigational Site, Boise, Idaho
  - 1245.25.10097 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1245.25.10116 Boehringer Ingelheim Investigational Site, Evansville, Indiana
  - 1245.25.10206 Boehringer Ingelheim Investigational Site, Valparaiso, Indiana
  - 1245.25.10021 Boehringer Ingelheim Investigational Site, Wichita, Kansas
  - 1245.25.10186 Boehringer Ingelheim Investigational Site, Lexington, Kentucky
  - 1245.25.10109 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 1245.25.10006 Boehringer Ingelheim Investigational Site, Madisonville, Kentucky
  - 1245.25.10005 Boehringer Ingelheim Investigational Site, Paducah, Kentucky
  - 1245.25.10020 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 1245.25.10012 Boehringer Ingelheim Investigational Site, Auburn, Maine
  - 1245.25.10041 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1245.25.10134 Boehringer Ingelheim Investigational Site, Hyattsville, Maryland
  - 1245.25.10210 Boehringer Ingelheim Investigational Site, Towson, Maryland
  - 1245.25.10064 Boehringer Ingelheim Investigational Site, Springfield, Massachusetts
  - 1245.25.10051 Boehringer Ingelheim Investigational Site, Watertown, Massachusetts
  - 1245.25.10071 Boehringer Ingelheim Investigational Site, Dearborn, Michigan
  - 1245.25.10013 Boehringer Ingelheim Investigational Site, Flint, Michigan
  - 1245.25.10107 Boehringer Ingelheim Investigational Site, Petoskey, Michigan
  - 1245.25.10030 Boehringer Ingelheim Investigational Site, Eagan, Minnesota
  - 1245.25.10028 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 1245.25.10176 Boehringer Ingelheim Investigational Site, Picayune, Mississippi
  - 1245.25.10011 Boehringer Ingelheim Investigational Site, Chesterfield, Missouri
  - 1245.25.10163 Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 1245.25.10148 Boehringer Ingelheim Investigational Site, Great Falls, Montana
  - 1245.25.10191 Boehringer Ingelheim Investigational Site, Great Falls, Montana
  - 1245.25.10034 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 1245.25.10014 Boehringer Ingelheim Investigational Site, Flemington, New Jersey
  - 1245.25.10145 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 1245.25.10180 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 1245.25.10131 Boehringer Ingelheim Investigational Site, Binghamton, New York
  - 1245.25.10029 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 1245.25.10142 Boehringer Ingelheim Investigational Site, Smithtown, New York
  - 1245.25.10096 Boehringer Ingelheim Investigational Site, Staten Island, New York
  - 1245.25.10196 Boehringer Ingelheim Investigational Site, Burlington, North Carolina
  - 1245.25.10207 Boehringer Ingelheim Investigational Site, Calabash, North Carolina
  - 1245.25.10053 Boehringer Ingelheim Investigational Site, Durham, North Carolina
  - 1245.25.10010 Boehringer Ingelheim Investigational Site, Greenville, North Carolina
  - 1245.25.10060 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1245.25.10086 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1245.25.10137 Boehringer Ingelheim Investigational Site, Dayton, Ohio
  - 1245.25.10138 Boehringer Ingelheim Investigational Site, Delaware, Ohio
  - 1245.25.10156 Boehringer Ingelheim Investigational Site, Kettering, Ohio
  - 1245.25.10091 Boehringer Ingelheim Investigational Site, Marion, Ohio
  - 1245.25.10192 Boehringer Ingelheim Investigational Site, Zanesville, Ohio
  - 1245.25.10114 Boehringer Ingelheim Investigational Site, Norman, Oklahoma
  - 1245.25.10082 Boehringer Ingelheim Investigational Site, Eugene, Oregon
  - 1245.25.10154 Boehringer Ingelheim Investigational Site, Clairton, Pennsylvania
  - 1245.25.10173 Boehringer Ingelheim Investigational Site, Clairton, Pennsylvania
  - 1245.25.10052 Boehringer Ingelheim Investigational Site, Feasterville-Trevose, Pennsylvania
  - 1245.25.10069 Boehringer Ingelheim Investigational Site, Fleetwood, Pennsylvania
  - 1245.25.10172 Boehringer Ingelheim Investigational Site, Greensburg, Pennsylvania
  - 1245.25.10050 Boehringer Ingelheim Investigational Site, Indiana, Pennsylvania
  - 1245.25.10009 Boehringer Ingelheim Investigational Site, Lansdale, Pennsylvania
  - 1245.25.10214 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1245.25.10149 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1245.25.10197 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1245.25.10159 Boehringer Ingelheim Investigational Site, Scottdale, Pennsylvania
  - 1245.25.10162 Boehringer Ingelheim Investigational Site, Tipton, Pennsylvania
  - 1245.25.10146 Boehringer Ingelheim Investigational Site, Uniontown, Pennsylvania
  - 1245.25.10077 Boehringer Ingelheim Investigational Site, Yardley, Pennsylvania
  - 1245.25.10070 Boehringer Ingelheim Investigational Site, Anderson, South Carolina
  - 1245.25.10044 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1245.25.10002 Boehringer Ingelheim Investigational Site, Greer, South Carolina
  - 1245.25.10132 Boehringer Ingelheim Investigational Site, Hodges, South Carolina
  - 1245.25.10140 Boehringer Ingelheim Investigational Site, Mt. Pleasant, South Carolina
  - 1245.25.10065 Boehringer Ingelheim Investigational Site, Myrtle Beach, South Carolina
  - 1245.25.10127 Boehringer Ingelheim Investigational Site, Myrtle Beach, South Carolina
  - 1245.25.10170 Boehringer Ingelheim Investigational Site, North Myrtle Beach, South Carolina
  - 1245.25.10129 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1245.25.10171 Boehringer Ingelheim Investigational Site, Union, South Carolina
  - 1245.25.10054 Boehringer Ingelheim Investigational Site, Bristol, Tennessee
  - 1245.25.10036 Boehringer Ingelheim Investigational Site, Chattanooga, Tennessee
  - 1245.25.10057 Boehringer Ingelheim Investigational Site, Chattanooga, Tennessee
  - 1245.25.10046 Boehringer Ingelheim Investigational Site, Kingsport, Tennessee
  - 1245.25.10143 Boehringer Ingelheim Investigational Site, Memphis, Tennessee
  - 1245.25.10075 Boehringer Ingelheim Investigational Site, Corpus Christi, Texas
  - 1245.25.10007 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1245.25.10026 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1245.25.10100 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1245.25.10165 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1245.25.10169 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 1245.25.10003 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1245.25.10125 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1245.25.10189 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1245.25.10119 Boehringer Ingelheim Investigational Site, Lubbock, Texas
  - 1245.25.10078 Boehringer Ingelheim Investigational Site, New Braunfels, Texas
  - 1245.25.10076 Boehringer Ingelheim Investigational Site, Odessa, Texas
  - 1245.25.10133 Boehringer Ingelheim Investigational Site, Pearland, Texas
  - 1245.25.10160 Boehringer Ingelheim Investigational Site, Plano, Texas
  - 1245.25.10177 Boehringer Ingelheim Investigational Site, Richardson, Texas
  - 1245.25.10049 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1245.25.10161 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1245.25.10185 Boehringer Ingelheim Investigational Site, Bountiful, Utah
  - 1245.25.10155 Boehringer Ingelheim Investigational Site, Draper, Utah
  - 1245.25.10079 Boehringer Ingelheim Investigational Site, Midvale, Utah
  - 1245.25.10080 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 1245.25.10087 Boehringer Ingelheim Investigational Site, South Ogden, Utah
  - 1245.25.10218 Boehringer Ingelheim Investigational Site, Burke, Virginia
  - 1245.25.10004 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
  - 1245.25.10111 Boehringer Ingelheim Investigational Site, South Chesterfield, Virginia
  - 1245.25.10115 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 1245.25.10216 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 1245.25.10017 Boehringer Ingelheim Investigational Site, Tacoma, Washington
  - 1245.25.10016 Boehringer Ingelheim Investigational Site, Walla Walla, Washington
  - 1245.25.10187 Boehringer Ingelheim Investigational Site, Charleston, West Virginia
  - 1245.25.10182 Boehringer Ingelheim Investigational Site, Morgantown, West Virginia
  - 1245.25.10098 Boehringer Ingelheim Investigational Site, Madison, Wisconsin
- Argentina (11):
  - 1245.25.54012 Boehringer Ingelheim Investigational Site, Buenos Aires
  - 1245.25.54001 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1245.25.54006 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1245.25.54013 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1245.25.54002 Boehringer Ingelheim Investigational Site, Córdoba
  - 1245.25.54003 Boehringer Ingelheim Investigational Site, Córdoba
  - 1245.25.54010 Boehringer Ingelheim Investigational Site, Córdoba
  - 1245.25.54011 Boehringer Ingelheim Investigational Site, Córdoba
  - 1245.25.54005 Boehringer Ingelheim Investigational Site, Parque Velez Sarfield
  - 1245.25.54008 Boehringer Ingelheim Investigational Site, Rosario
  - 1245.25.54009 Boehringer Ingelheim Investigational Site, Rosario
- Australia (3):
  - 1245.25.61003 Boehringer Ingelheim Investigational Site, Herston, Queensland
  - 1245.25.61001 Boehringer Ingelheim Investigational Site, Ashford, South Australia
  - 1245.25.61002 Boehringer Ingelheim Investigational Site, Fullarton, South Australia
- Austria (10):
  - 1245.25.43008 Boehringer Ingelheim Investigational Site, Feldkirch
  - 1245.25.43006 Boehringer Ingelheim Investigational Site, Graz
  - 1245.25.43016 Boehringer Ingelheim Investigational Site, Innsbruck
  - 1245.25.43005 Boehringer Ingelheim Investigational Site, Salzburg
  - 1245.25.43015 Boehringer Ingelheim Investigational Site, St. Stefan
  - 1245.25.43001 Boehringer Ingelheim Investigational Site, Vienna
  - 1245.25.43007 Boehringer Ingelheim Investigational Site, Vienna
  - 1245.25.43009 Boehringer Ingelheim Investigational Site, Vienna
  - 1245.25.43010 Boehringer Ingelheim Investigational Site, Vienna
  - 1245.25.43013 Boehringer Ingelheim Investigational Site, Vienna
- Belgium (16):
  - 1245.25.32010 Boehringer Ingelheim Investigational Site, Bonheiden
  - 1245.25.32008 Boehringer Ingelheim Investigational Site, Brussels
  - 1245.25.32011 Boehringer Ingelheim Investigational Site, Brussels
  - 1245.25.32030 Boehringer Ingelheim Investigational Site, Brussels
  - 1245.25.32003 Boehringer Ingelheim Investigational Site, De Pinte
  - 1245.25.32002 Boehringer Ingelheim Investigational Site, Edegem
  - 1245.25.32004 Boehringer Ingelheim Investigational Site, Genk
  - 1245.25.32029 Boehringer Ingelheim Investigational Site, Halen
  - 1245.25.32009 Boehringer Ingelheim Investigational Site, Hasselt
  - 1245.25.32007 Boehringer Ingelheim Investigational Site, Huy
  - 1245.25.32013 Boehringer Ingelheim Investigational Site, La Louvière
  - 1245.25.32012 Boehringer Ingelheim Investigational Site, Leuven
  - 1245.25.32001 Boehringer Ingelheim Investigational Site, Liège
  - 1245.25.32028 Boehringer Ingelheim Investigational Site, Liège
  - 1245.25.32005 Boehringer Ingelheim Investigational Site, Massemen-Wetteren
  - 1245.25.32014 Boehringer Ingelheim Investigational Site, Oostham
- Brazil (25):
  - 1245.25.55014 Boehringer Ingelheim Investigational Site, Belém
  - 1245.25.55019 Boehringer Ingelheim Investigational Site, Belo Horizonte
  - 1245.25.55007 Boehringer Ingelheim Investigational Site, Boqueirão
  - 1245.25.55015 Boehringer Ingelheim Investigational Site, Brasília
  - 1245.25.55027 Boehringer Ingelheim Investigational Site, Campinas
  - 1245.25.55028 Boehringer Ingelheim Investigational Site, Campinas
  - 1245.25.55025 Boehringer Ingelheim Investigational Site, Curitiba
  - 1245.25.55026 Boehringer Ingelheim Investigational Site, Fortaleza
  - 1245.25.55009 Boehringer Ingelheim Investigational Site, Goiânia
  - 1245.25.55002 Boehringer Ingelheim Investigational Site, Higienópolis
  - 1245.25.55022 Boehringer Ingelheim Investigational Site, Maringá
  - 1245.25.55017 Boehringer Ingelheim Investigational Site, Marília
  - 1245.25.55008 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 1245.25.55016 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 1245.25.55020 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 1245.25.55012 Boehringer Ingelheim Investigational Site, Ribeirão Preto
  - 1245.25.55013 Boehringer Ingelheim Investigational Site, São José do Rio Preto
  - 1245.25.55004 Boehringer Ingelheim Investigational Site, São Paulo
  - 1245.25.55010 Boehringer Ingelheim Investigational Site, São Paulo
  - 1245.25.55018 Boehringer Ingelheim Investigational Site, São Paulo
  - 1245.25.55023 Boehringer Ingelheim Investigational Site, São Paulo
  - 1245.25.55006 Boehringer Ingelheim Investigational Site, Vila Albuquerque
  - 1245.25.55003 Boehringer Ingelheim Investigational Site, Vila Clementino
  - 1245.25.55005 Boehringer Ingelheim Investigational Site, Vila Leopoldina
  - 1245.25.55001 Boehringer Ingelheim Investigational Site, Villa Clementino
- Canada (13):
  - 1245.25.20047 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1245.25.20048 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 1245.25.20026 Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - 1245.25.20045 Boehringer Ingelheim Investigational Site, Brampton, Ontario
  - 1245.25.20042 Boehringer Ingelheim Investigational Site, Burlington, Ontario
  - 1245.25.20009 Boehringer Ingelheim Investigational Site, Newmarket, Ontario
  - 1245.25.20044 Boehringer Ingelheim Investigational Site, Niagara Falls, Ontario
  - 1245.25.20013 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1245.25.20049 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1245.25.20050 Boehringer Ingelheim Investigational Site, Gatineau, Quebec
  - 1245.25.20043 Boehringer Ingelheim Investigational Site, Longueuil, Quebec
  - 1245.25.20046 Boehringer Ingelheim Investigational Site, Longueuil, Quebec
  - 1245.25.20041 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- Colombia (7):
  - 1245.25.57010 Boehringer Ingelheim Investigational Site, Armenia
  - 1245.25.57004 Boehringer Ingelheim Investigational Site, Barranquilla
  - 1245.25.57001 Boehringer Ingelheim Investigational Site, Bogotá
  - 1245.25.57003 Boehringer Ingelheim Investigational Site, Bogotá
  - 1245.25.57011 Boehringer Ingelheim Investigational Site, Bogotá
  - 1245.25.57006 Boehringer Ingelheim Investigational Site, Floridablanca
  - 1245.25.57009 Boehringer Ingelheim Investigational Site, Medellín
- Croatia (6):
  - 1245.25.71005 Boehringer Ingelheim Investigational Site, Karlovac
  - 1245.25.71001 Boehringer Ingelheim Investigational Site, Krapinske Toplice
  - 1245.25.71006 Boehringer Ingelheim Investigational Site, Osijek
  - 1245.25.71003 Boehringer Ingelheim Investigational Site, Rijeka
  - 1245.25.71002 Boehringer Ingelheim Investigational Site, Zagreb
  - 1245.25.71004 Boehringer Ingelheim Investigational Site, Zagreb
- Czechia (4):
  - 1245.25.42020 Boehringer Ingelheim Investigational Site, Brno
  - 1245.25.42018 Boehringer Ingelheim Investigational Site, Jindřichův Hradec
  - 1245.25.42015 Boehringer Ingelheim Investigational Site, Prague
  - 1245.25.42019 Boehringer Ingelheim Investigational Site, Ústí nad Labem
- Denmark (6):
  - 1245.25.45007 Boehringer Ingelheim Investigational Site, Elsinore
  - 1245.25.45006 Boehringer Ingelheim Investigational Site, Frederiksberg
  - 1245.25.45003 Boehringer Ingelheim Investigational Site, Gentofte Municipality
  - 1245.25.45002 Boehringer Ingelheim Investigational Site, København NV
  - 1245.25.45004 Boehringer Ingelheim Investigational Site, Randers NØ
  - 1245.25.45005 Boehringer Ingelheim Investigational Site, Slagelse
- Estonia (5):
  - 1245.25.37002 Boehringer Ingelheim Investigational Site, Tallinn
  - 1245.25.37003 Boehringer Ingelheim Investigational Site, Tallinn
  - 1245.25.37005 Boehringer Ingelheim Investigational Site, Tallinn
  - 1245.25.37001 Boehringer Ingelheim Investigational Site, Tartu
  - 1245.25.37004 Boehringer Ingelheim Investigational Site, Tartu
- France (16):
  - 1245.25.33022 Boehringer Ingelheim Investigational Site, Amiens
  - 1245.25.33033 Boehringer Ingelheim Investigational Site, Angers
  - 1245.25.33034 Boehringer Ingelheim Investigational Site, Angers
  - 1245.25.33030 Boehringer Ingelheim Investigational Site, Bourg Des Cptes
  - 1245.25.33023 Boehringer Ingelheim Investigational Site, Corbeil-Essonnes
  - 1245.25.33024 Boehringer Ingelheim Investigational Site, Derval
  - 1245.25.33029 Boehringer Ingelheim Investigational Site, Equeurdreville Haineville
  - 1245.25.33027 Boehringer Ingelheim Investigational Site, Fleury-sur-Orne
  - 1245.25.33021 Boehringer Ingelheim Investigational Site, Grenoble
  - 1245.25.33003 Boehringer Ingelheim Investigational Site, La Rochelle
  - 1245.25.33032 Boehringer Ingelheim Investigational Site, Le Creusot
  - 1245.25.33004 Boehringer Ingelheim Investigational Site, Narbonne
  - 1245.25.33047 Boehringer Ingelheim Investigational Site, Pessac
  - 1245.25.33046 Boehringer Ingelheim Investigational Site, Poitiers
  - 1245.25.33025 Boehringer Ingelheim Investigational Site, Saint Priez En Jarez
  - 1245.25.33035 Boehringer Ingelheim Investigational Site, Tours
- Georgia (8):
  - 1245.25.99001 Boehringer Ingelheim Investigational Site, Batumi
  - 1245.25.99003 Boehringer Ingelheim Investigational Site, Kutaisi
  - 1245.25.99002 Boehringer Ingelheim Investigational Site, Tbilisi
  - 1245.25.99004 Boehringer Ingelheim Investigational Site, Tbilisi
  - 1245.25.99005 Boehringer Ingelheim Investigational Site, Tbilisi
  - 1245.25.99006 Boehringer Ingelheim Investigational Site, Tbilisi
  - 1245.25.99007 Boehringer Ingelheim Investigational Site, Tbilisi
  - 1245.25.99008 Boehringer Ingelheim Investigational Site, Tbilisi
- Greece (8):
  - 1245.25.30002 Boehringer Ingelheim Investigational Site, Athens
  - 1245.25.30003 Boehringer Ingelheim Investigational Site, Athens
  - 1245.25.30004 Boehringer Ingelheim Investigational Site, Athens
  - 1245.25.30007 Boehringer Ingelheim Investigational Site, Athens
  - 1245.25.30005 Boehringer Ingelheim Investigational Site, Larissa
  - 1245.25.30001 Boehringer Ingelheim Investigational Site, Nikaia
  - 1245.25.30006 Boehringer Ingelheim Investigational Site, Thessaloniki
  - 1245.25.30008 Boehringer Ingelheim Investigational Site, Thessaloniki
- Hong Kong (4):
  - 1245.25.85201 Boehringer Ingelheim Investigational Site, Hong Kong
  - 1245.25.85205 Boehringer Ingelheim Investigational Site, Hong Kong
  - 1245.25.85207 Boehringer Ingelheim Investigational Site, Hong Kong
  - 1245.25.85208 Boehringer Ingelheim Investigational Site, Hong Kong
- Hungary (8):
  - 1245.25.36002 Boehringer Ingelheim Investigational Site, Budapest
  - 1245.25.36004 Boehringer Ingelheim Investigational Site, Budapest
  - 1245.25.36008 Boehringer Ingelheim Investigational Site, Budapest
  - 1245.25.36006 Boehringer Ingelheim Investigational Site, Dunaújváros
  - 1245.25.36001 Boehringer Ingelheim Investigational Site, Gyula
  - 1245.25.36010 Boehringer Ingelheim Investigational Site, Kisvárda
  - 1245.25.36003 Boehringer Ingelheim Investigational Site, Szekszárd
  - 1245.25.36011 Boehringer Ingelheim Investigational Site, Szikszó
- India (18):
  - 1245.25.91307 Boehringer Ingelheim Investigational Site, Ahmedabad
  - 1245.25.91302 Boehringer Ingelheim Investigational Site, Bangalore
  - 1245.25.91317 Boehringer Ingelheim Investigational Site, Bangalore
  - 1245.25.91319 Boehringer Ingelheim Investigational Site, Bangalore
  - 1245.25.91320 Boehringer Ingelheim Investigational Site, Bangalore
  - 1245.25.91303 Boehringer Ingelheim Investigational Site, Chennai
  - 1245.25.91311 Boehringer Ingelheim Investigational Site, Hyderabad
  - 1245.25.91318 Boehringer Ingelheim Investigational Site, Indore
  - 1245.25.91305 Boehringer Ingelheim Investigational Site, Jaipur
  - 1245.25.91309 Boehringer Ingelheim Investigational Site, Jalandhar
  - 1245.25.91315 Boehringer Ingelheim Investigational Site, Kochi
  - 1245.25.91313 Boehringer Ingelheim Investigational Site, Nagpur
  - 1245.25.91324 Boehringer Ingelheim Investigational Site, Nagpur
  - 1245.25.91301 Boehringer Ingelheim Investigational Site, Nashik, Maharashtra
  - 1245.25.91308 Boehringer Ingelheim Investigational Site, Pune
  - 1245.25.91316 Boehringer Ingelheim Investigational Site, Secunderabad
  - 1245.25.91321 Boehringer Ingelheim Investigational Site, Varanasi
  - 1245.25.91314 Boehringer Ingelheim Investigational Site, Vijaywada
- Indonesia (8):
  - 1245.25.62006 Boehringer Ingelheim Investigational Site, Denpasar
  - 1245.25.62009 Boehringer Ingelheim Investigational Site, Depok
  - 1245.25.62002 Boehringer Ingelheim Investigational Site, Jakarta
  - 1245.25.62008 Boehringer Ingelheim Investigational Site, Jakarta
  - 1245.25.62010 Boehringer Ingelheim Investigational Site, Jakarta
  - 1245.25.62004 Boehringer Ingelheim Investigational Site, Malang
  - 1245.25.62003 Boehringer Ingelheim Investigational Site, Surabaya
  - 1245.25.62001 Boehringer Ingelheim Investigational Site, Yogyakarta
- Israel (7):
  - 1245.25.97003 Boehringer Ingelheim Investigational Site, Afula
  - 1245.25.97006 Boehringer Ingelheim Investigational Site, Hadera
  - 1245.25.97008 Boehringer Ingelheim Investigational Site, Haifa
  - 1245.25.97009 Boehringer Ingelheim Investigational Site, Holon
  - 1245.25.97005 Boehringer Ingelheim Investigational Site, Nahariya
  - 1245.25.97001 Boehringer Ingelheim Investigational Site, Safed
  - 1245.25.97002 Boehringer Ingelheim Investigational Site, Ẕerifin
- Italy (15):
  - 1245.25.39007 Boehringer Ingelheim Investigational Site, Bologna
  - 1245.25.39002 Boehringer Ingelheim Investigational Site, Campobasso
  - 1245.25.39008 Boehringer Ingelheim Investigational Site, Catanzaro
  - 1245.25.39010 Boehringer Ingelheim Investigational Site, Chieti
  - 1245.25.39024 Boehringer Ingelheim Investigational Site, Ferrara
  - 1245.25.39009 Boehringer Ingelheim Investigational Site, Florence
  - 1245.25.39005 Boehringer Ingelheim Investigational Site, Foggia
  - 1245.25.39004 Boehringer Ingelheim Investigational Site, Napoli
  - 1245.25.39006 Boehringer Ingelheim Investigational Site, Padua
  - 1245.25.39001 Boehringer Ingelheim Investigational Site, Pisa
  - 1245.25.39003 Boehringer Ingelheim Investigational Site, Roma
  - 1245.25.39011 Boehringer Ingelheim Investigational Site, Roma
  - 1245.25.39012 Boehringer Ingelheim Investigational Site, Roma
  - 1245.25.39014 Boehringer Ingelheim Investigational Site, Roma
  - 1245.25.39013 Boehringer Ingelheim Investigational Site, Venezia
- Japan (14):
  - 1245.25.81008 Boehringer Ingelheim Investigational Site, Chuo-ku, Tokyo
  - 1245.25.81010 Boehringer Ingelheim Investigational Site, Gifushi, Gifu
  - 1245.25.81002 Boehringer Ingelheim Investigational Site, Hanyushi, Saitama
  - 1245.25.81013 Boehringer Ingelheim Investigational Site, Kamigyo-ku, Kyotoshi, Kyoto
  - 1245.25.81003 Boehringer Ingelheim Investigational Site, Kishiwadashi. Osaka
  - 1245.25.81012 Boehringer Ingelheim Investigational Site, Kita-ku, Nagoyashi, Aichi
  - 1245.25.81014 Boehringer Ingelheim Investigational Site, Kumamoto-shi, Kumamoto
  - 1245.25.81001 Boehringer Ingelheim Investigational Site, Matsudoshi, Chiba
  - 1245.25.81006 Boehringer Ingelheim Investigational Site, Mitoshi, Ibaraki
  - 1245.25.81005 Boehringer Ingelheim Investigational Site, Nishi-ku, Sapporoshi, Hokkaido
  - 1245.25.81007 Boehringer Ingelheim Investigational Site, Nodashi, Chiba
  - 1245.25.81004 Boehringer Ingelheim Investigational Site, Shimajiri-gun,Okinawa
  - 1245.25.81009 Boehringer Ingelheim Investigational Site, Toyamashi, Toyama
  - 1245.25.81015 Boehringer Ingelheim Investigational Site, Toyoakeshi, Aichi
- Malaysia (10):
  - 1245.25.60019 Boehringer Ingelheim Investigational Site, Johor Bahru
  - 1245.25.60020 Boehringer Ingelheim Investigational Site, Kedah
  - 1245.25.60013 Boehringer Ingelheim Investigational Site, Kelantan
  - 1245.25.60015 Boehringer Ingelheim Investigational Site, Kota Kinabalu
  - 1245.25.60012 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 1245.25.60017 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 1245.25.60004 Boehringer Ingelheim Investigational Site, Kuala Pahang
  - 1245.25.60016 Boehringer Ingelheim Investigational Site, Kuala Selangor
  - 1245.25.60021 Boehringer Ingelheim Investigational Site, Kuala Selangor
  - 1245.25.60018 Boehringer Ingelheim Investigational Site, Selangor Darul Ehsan
- Mexico (7):
  - 1245.25.52009 Boehringer Ingelheim Investigational Site, Colonia Americana
  - 1245.25.52007 Boehringer Ingelheim Investigational Site, Distrito Federal
  - 1245.25.52013 Boehringer Ingelheim Investigational Site, Ladrón de Guevara
  - 1245.25.52010 Boehringer Ingelheim Investigational Site, Los Robles
  - 1245.25.52001 Boehringer Ingelheim Investigational Site, Monterrey
  - 1245.25.52011 Boehringer Ingelheim Investigational Site, Reforma Social
  - 1245.25.52012 Boehringer Ingelheim Investigational Site, San Lucas Tepetlcalco
- Netherlands (20):
  - 1245.25.31015 Boehringer Ingelheim Investigational Site, Amersfoort
  - 1245.25.31013 Boehringer Ingelheim Investigational Site, Apeldoorn
  - 1245.25.31036 Boehringer Ingelheim Investigational Site, Baarle-Nassau
  - 1245.25.31032 Boehringer Ingelheim Investigational Site, Delft
  - 1245.25.31026 Boehringer Ingelheim Investigational Site, Den Helder
  - 1245.25.31012 Boehringer Ingelheim Investigational Site, Geleen
  - 1245.25.31017 Boehringer Ingelheim Investigational Site, Hardenberg
  - 1245.25.31035 Boehringer Ingelheim Investigational Site, Heerlen
  - 1245.25.31011 Boehringer Ingelheim Investigational Site, Hoogeveen
  - 1245.25.31029 Boehringer Ingelheim Investigational Site, Hoogezand
  - 1245.25.31023 Boehringer Ingelheim Investigational Site, Hoogwoud
  - 1245.25.31009 Boehringer Ingelheim Investigational Site, Maastricht
  - 1245.25.31031 Boehringer Ingelheim Investigational Site, Meppel
  - 1245.25.31024 Boehringer Ingelheim Investigational Site, Nijverdal
  - 1245.25.31014 Boehringer Ingelheim Investigational Site, Rotterdam
  - 1245.25.31033 Boehringer Ingelheim Investigational Site, Rotterdam
  - 1245.25.31030 Boehringer Ingelheim Investigational Site, Schiedam
  - 1245.25.31002 Boehringer Ingelheim Investigational Site, Utrecht
  - 1245.25.31028 Boehringer Ingelheim Investigational Site, Wildervank
  - 1245.25.31034 Boehringer Ingelheim Investigational Site, Zutphen
- New Zealand (3):
  - 1245.25.64004 Boehringer Ingelheim Investigational Site, Christchurch
  - 1245.25.64001 Boehringer Ingelheim Investigational Site, Grafton / Auckland
  - 1245.25.64003 Boehringer Ingelheim Investigational Site, Wellington
- Norway (8):
  - 1245.25.47002 Boehringer Ingelheim Investigational Site, Fornebu
  - 1245.25.47004 Boehringer Ingelheim Investigational Site, Gjøvik
  - 1245.25.47009 Boehringer Ingelheim Investigational Site, Kløfta
  - 1245.25.47008 Boehringer Ingelheim Investigational Site, Kongsvinger
  - 1245.25.47001 Boehringer Ingelheim Investigational Site, Oslo
  - 1245.25.47006 Boehringer Ingelheim Investigational Site, Oslo
  - 1245.25.47007 Boehringer Ingelheim Investigational Site, Trondheim
  - 1245.25.47005 Boehringer Ingelheim Investigational Site, Tynset
- Peru (11):
  - 1245.25.51001 Boehringer Ingelheim Investigational Site, Arequipa
  - 1245.25.51008 Boehringer Ingelheim Investigational Site, Arequipa
  - 1245.25.51002 Boehringer Ingelheim Investigational Site, Bellavista
  - 1245.25.51004 Boehringer Ingelheim Investigational Site, El Agustino
  - 1245.25.51006 Boehringer Ingelheim Investigational Site, Ica
  - 1245.25.51003 Boehringer Ingelheim Investigational Site, Jesus Maria
  - 1245.25.51007 Boehringer Ingelheim Investigational Site, Lima
  - 1245.25.51009 Boehringer Ingelheim Investigational Site, Lima
  - 1245.25.51010 Boehringer Ingelheim Investigational Site, Lima
  - 1245.25.51011 Boehringer Ingelheim Investigational Site, Lima
  - 1245.25.51005 Boehringer Ingelheim Investigational Site, Miraflores
- Philippines (10):
  - 1245.25.63016 Boehringer Ingelheim Investigational Site, Cavite City
  - 1245.25.63002 Boehringer Ingelheim Investigational Site, Cebu
  - 1245.25.63003 Boehringer Ingelheim Investigational Site, Davao City
  - 1245.25.63020 Boehringer Ingelheim Investigational Site, Jaro Iloilo City
  - 1245.25.63001 Boehringer Ingelheim Investigational Site, Manila
  - 1245.25.63004 Boehringer Ingelheim Investigational Site, Manila
  - 1245.25.63018 Boehringer Ingelheim Investigational Site, Manila
  - 1245.25.63009 Boehringer Ingelheim Investigational Site, Marikina City
  - 1245.25.63021 Boehringer Ingelheim Investigational Site, Marikina City
  - 1245.25.63019 Boehringer Ingelheim Investigational Site, Tarlac City
- Poland (11):
  - 1245.25.48013 Boehringer Ingelheim Investigational Site, Gdansk
  - 1245.25.48004 Boehringer Ingelheim Investigational Site, Lodz
  - 1245.25.48009 Boehringer Ingelheim Investigational Site, Lodz
  - 1245.25.48010 Boehringer Ingelheim Investigational Site, Lodz
  - 1245.25.48001 Boehringer Ingelheim Investigational Site, Lublin
  - 1245.25.48014 Boehringer Ingelheim Investigational Site, Oświęcim
  - 1245.25.48002 Boehringer Ingelheim Investigational Site, Poznan
  - 1245.25.48008 Boehringer Ingelheim Investigational Site, Puławy
  - 1245.25.48007 Boehringer Ingelheim Investigational Site, Ruda Śląska
  - 1245.25.48005 Boehringer Ingelheim Investigational Site, Torun
  - 1245.25.48011 Boehringer Ingelheim Investigational Site, Torun
- Portugal (14):
  - 1245.25.35006 Boehringer Ingelheim Investigational Site, Amadora
  - 1245.25.35004 Boehringer Ingelheim Investigational Site, Coimbra
  - 1245.25.35018 Boehringer Ingelheim Investigational Site, Faro
  - 1245.25.35021 Boehringer Ingelheim Investigational Site, Funchal
  - 1245.25.35008 Boehringer Ingelheim Investigational Site, Leiria
  - 1245.25.35001 Boehringer Ingelheim Investigational Site, Lisbon
  - 1245.25.35002 Boehringer Ingelheim Investigational Site, Lisbon
  - 1245.25.35015 Boehringer Ingelheim Investigational Site, Lisbon
  - 1245.25.35017 Boehringer Ingelheim Investigational Site, Lisbon
  - 1245.25.35011 Boehringer Ingelheim Investigational Site, Porto
  - 1245.25.35005 Boehringer Ingelheim Investigational Site, Santiago do Cacém
  - 1245.25.35020 Boehringer Ingelheim Investigational Site, Torres Novas
  - 1245.25.35014 Boehringer Ingelheim Investigational Site, Viana do Castelo
  - 1245.25.35019 Boehringer Ingelheim Investigational Site, Vila Nova de Gaia
- Romania (9):
  - 1245.25.40008 Boehringer Ingelheim Investigational Site, Alba Iulia
  - 1245.25.40011 Boehringer Ingelheim Investigational Site, Baia Mare Maramures
  - 1245.25.40003 Boehringer Ingelheim Investigational Site, Bucharest
  - 1245.25.40007 Boehringer Ingelheim Investigational Site, Bucharest
  - 1245.25.40005 Boehringer Ingelheim Investigational Site, Constanța
  - 1245.25.40002 Boehringer Ingelheim Investigational Site, Craiova
  - 1245.25.40006 Boehringer Ingelheim Investigational Site, Craiova
  - 1245.25.40009 Boehringer Ingelheim Investigational Site, Oradea
  - 1245.25.40010 Boehringer Ingelheim Investigational Site, Târgu Mureş
- Russia (25):
  - 1245.25.70019 Boehringer Ingelheim Investigational Site, Barnaul
  - 1245.25.70015 Boehringer Ingelheim Investigational Site, Kemerovo
  - 1245.25.70020 Boehringer Ingelheim Investigational Site, Kemerovo
  - 1245.25.70003 Boehringer Ingelheim Investigational Site, Moscow
  - 1245.25.70009 Boehringer Ingelheim Investigational Site, Moscow
  - 1245.25.70011 Boehringer Ingelheim Investigational Site, Moscow
  - 1245.25.70016 Boehringer Ingelheim Investigational Site, Moscow
  - 1245.25.70021 Boehringer Ingelheim Investigational Site, Moscow
  - 1245.25.70022 Boehringer Ingelheim Investigational Site, Moscow
  - 1245.25.70014 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 1245.25.70018 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 1245.25.70024 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 1245.25.70028 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 1245.25.70001 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1245.25.70004 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1245.25.70005 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1245.25.70006 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1245.25.70013 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1245.25.70017 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1245.25.70023 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1245.25.70025 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1245.25.70026 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1245.25.70027 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1245.25.70002 Boehringer Ingelheim Investigational Site, Vsevolozhsk
  - 1245.25.70029 Boehringer Ingelheim Investigational Site, Yaroslavl
- Singapore (3):
  - 1245.25.65001 Boehringer Ingelheim Investigational Site, Singapore
  - 1245.25.65003 Boehringer Ingelheim Investigational Site, Singapore
  - 1245.25.65004 Boehringer Ingelheim Investigational Site, Singapore
- South Africa (21):
  - 1245.25.76007 Boehringer Ingelheim Investigational Site, Alberton
  - 1245.25.76002 Boehringer Ingelheim Investigational Site, Bellville
  - 1245.25.76009 Boehringer Ingelheim Investigational Site, Bloemfontein
  - 1245.25.76014 Boehringer Ingelheim Investigational Site, Cape Town
  - 1245.25.76020 Boehringer Ingelheim Investigational Site, Cape Town
  - 1245.25.76022 Boehringer Ingelheim Investigational Site, Chatsworth Unit 10
  - 1245.25.76013 Boehringer Ingelheim Investigational Site, Durban
  - 1245.25.76016 Boehringer Ingelheim Investigational Site, Durban
  - 1245.25.76019 Boehringer Ingelheim Investigational Site, Durban
  - 1245.25.76003 Boehringer Ingelheim Investigational Site, Goodwood
  - 1245.25.76001 Boehringer Ingelheim Investigational Site, Houghton Estate
  - 1245.25.76021 Boehringer Ingelheim Investigational Site, Kempton Park
  - 1245.25.76017 Boehringer Ingelheim Investigational Site, Krugersdorp
  - 1245.25.76004 Boehringer Ingelheim Investigational Site, Newtown
  - 1245.25.76006 Boehringer Ingelheim Investigational Site, Paarl
  - 1245.25.76005 Boehringer Ingelheim Investigational Site, Parow
  - 1245.25.76018 Boehringer Ingelheim Investigational Site, Port Elizabeth
  - 1245.25.76015 Boehringer Ingelheim Investigational Site, Somerset West
  - 1245.25.76012 Boehringer Ingelheim Investigational Site, Sydenham
  - 1245.25.76008 Boehringer Ingelheim Investigational Site, Tongaat
  - 1245.25.76023 Boehringer Ingelheim Investigational Site, Worcester
- South Korea (17):
  - 1245.25.82030 Boehringer Ingelheim Investigational Site, Busan
  - 1245.25.82018 Boehringer Ingelheim Investigational Site, Daegu
  - 1245.25.82021 Boehringer Ingelheim Investigational Site, Daejeon
  - 1245.25.82031 Boehringer Ingelheim Investigational Site, Daejoen
  - 1245.25.82027 Boehringer Ingelheim Investigational Site, Goyang
  - 1245.25.82022 Boehringer Ingelheim Investigational Site, Gwangju
  - 1245.25.82029 Boehringer Ingelheim Investigational Site, Incheon
  - 1245.25.82017 Boehringer Ingelheim Investigational Site, Pusan
  - 1245.25.82015 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.25.82016 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.25.82019 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.25.82020 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.25.82023 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.25.82024 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.25.82025 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.25.82026 Boehringer Ingelheim Investigational Site, Suwon
  - 1245.25.82028 Boehringer Ingelheim Investigational Site, Wŏnju
- Spain (23):
  - 1245.25.34025 Boehringer Ingelheim Investigational Site, Alcorcon (Madrid)
  - 1245.25.34048 Boehringer Ingelheim Investigational Site, Alicante
  - 1245.25.34050 Boehringer Ingelheim Investigational Site, Alzira
  - 1245.25.34039 Boehringer Ingelheim Investigational Site, Ávila
  - 1245.25.34040 Boehringer Ingelheim Investigational Site, Badía Del Vallès - Barcelona
  - 1245.25.34029 Boehringer Ingelheim Investigational Site, Barcelona
  - 1245.25.34030 Boehringer Ingelheim Investigational Site, Barcelona
  - 1245.25.34049 Boehringer Ingelheim Investigational Site, Barcelona
  - 1245.25.34031 Boehringer Ingelheim Investigational Site, Granada
  - 1245.25.34024 Boehringer Ingelheim Investigational Site, Leganes (Madrid)
  - 1245.25.34013 Boehringer Ingelheim Investigational Site, Madrid
  - 1245.25.34023 Boehringer Ingelheim Investigational Site, Madrid
  - 1245.25.34026 Boehringer Ingelheim Investigational Site, Madrid
  - 1245.25.34028 Boehringer Ingelheim Investigational Site, Madrid
  - 1245.25.34033 Boehringer Ingelheim Investigational Site, Madrid
  - 1245.25.34036 Boehringer Ingelheim Investigational Site, Madrid
  - 1245.25.34038 Boehringer Ingelheim Investigational Site, Madrid
  - 1245.25.34022 Boehringer Ingelheim Investigational Site, Mahadahonda (Madrid)
  - 1245.25.34047 Boehringer Ingelheim Investigational Site, Palma de Mallorca
  - 1245.25.34034 Boehringer Ingelheim Investigational Site, Sabadell (Barcelona)
  - 1245.25.34027 Boehringer Ingelheim Investigational Site, Salamanca
  - 1245.25.34037 Boehringer Ingelheim Investigational Site, Santa Cruz de Tenerife
  - 1245.25.34046 Boehringer Ingelheim Investigational Site, Segovia
- Sri Lanka (6):
  - 1245.25.94002 Boehringer Ingelheim Investigational Site, Colombo
  - 1245.25.94005 Boehringer Ingelheim Investigational Site, Kalubowila
  - 1245.25.94004 Boehringer Ingelheim Investigational Site, Kandy
  - 1245.25.94006 Boehringer Ingelheim Investigational Site, Kandy
  - 1245.25.94001 Boehringer Ingelheim Investigational Site, Nugegoda
  - 1245.25.94003 Boehringer Ingelheim Investigational Site, Ragama
- Taiwan (10):
  - 1245.25.88022 Boehringer Ingelheim Investigational Site, Hualien City
  - 1245.25.88010 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1245.25.88019 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1245.25.88009 Boehringer Ingelheim Investigational Site, Taichung
  - 1245.25.88020 Boehringer Ingelheim Investigational Site, Taichung
  - 1245.25.88018 Boehringer Ingelheim Investigational Site, Tainan
  - 1245.25.88015 Boehringer Ingelheim Investigational Site, Taipei
  - 1245.25.88016 Boehringer Ingelheim Investigational Site, Taipei
  - 1245.25.88023 Boehringer Ingelheim Investigational Site, Tamsui, Taipei County
  - 1245.25.88017 Boehringer Ingelheim Investigational Site, Taoyuan District
- Thailand (6):
  - 1245.25.66006 Boehringer Ingelheim Investigational Site, Bangkok
  - 1245.25.66007 Boehringer Ingelheim Investigational Site, Bangkok
  - 1245.25.66009 Boehringer Ingelheim Investigational Site, Chiang Mai
  - 1245.25.66004 Boehringer Ingelheim Investigational Site, Muang District
  - 1245.25.66010 Boehringer Ingelheim Investigational Site, Nakhonratchasima
  - 1245.25.66011 Boehringer Ingelheim Investigational Site, Pathum Tani
- Ukraine (7):
  - 1245.25.75001 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1245.25.75008 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1245.25.75009 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1245.25.75011 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1245.25.75007 Boehringer Ingelheim Investigational Site, Kiev
  - 1245.25.75012 Boehringer Ingelheim Investigational Site, Kiev
  - 1245.25.75010 Boehringer Ingelheim Investigational Site, Odesa
- United Kingdom (12):
  - 1245.25.44045 Boehringer Ingelheim Investigational Site, Airdrie
  - 1245.25.44020 Boehringer Ingelheim Investigational Site, Ashford
  - 1245.25.44013 Boehringer Ingelheim Investigational Site, Blackpool
  - 1245.25.44014 Boehringer Ingelheim Investigational Site, Bolton
  - 1245.25.44021 Boehringer Ingelheim Investigational Site, Bradford-on-Avon
  - 1245.25.44002 Boehringer Ingelheim Investigational Site, Dumfries
  - 1245.25.44009 Boehringer Ingelheim Investigational Site, Dundee
  - 1245.25.44005 Boehringer Ingelheim Investigational Site, Edinburgh
  - 1245.25.44004 Boehringer Ingelheim Investigational Site, Fowey
  - 1245.25.44001 Boehringer Ingelheim Investigational Site, Frome
  - 1245.25.44003 Boehringer Ingelheim Investigational Site, Inverness
  - 1245.25.44044 Boehringer Ingelheim Investigational Site, Wishaw

REFERENCES:
- [Derived] Odutayo A, Zinman B, Wanner C, Zwiener I, Lund SS, Hantel S, Fitchett D, Udell JA; EMPA-REG OUTCOME Trial Investigators. Effect of Qualifying Atherosclerotic Cardiovascular Disease Diagnosis Proximity on Cardiovascular Risk and Benefit of Empagliflozin in the EMPA-REG OUTCOME Trial. CJC Open. 2024 Feb 9;6(7):868-875. doi: 10.1016/j.cjco.2024.01.013. eCollection 2024 Jul. PMID 39026628
- [Derived] Fitchett D, Zinman B, Inzucchi SE, Wanner C, Anker SD, Pocock S, Mattheus M, Vedin O, Lund SS. Effect of empagliflozin on total myocardial infarction events by type and additional coronary outcomes: insights from the randomized EMPA-REG OUTCOME trial. Cardiovasc Diabetol. 2024 Jul 11;23(1):248. doi: 10.1186/s12933-024-02328-6. PMID 38992713
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Hadjadj S, Cooper ME, Steubl D, Petrini M, Hantel S, Mattheus M, Wanner C, Thomas MC. Empagliflozin and Rapid Kidney Function Decline Incidence in Type 2 Diabetes: An Exploratory Analysis From the EMPA-REG OUTCOME Trial. Kidney Med. 2023 Dec 18;6(3):100783. doi: 10.1016/j.xkme.2023.100783. eCollection 2024 Mar. PMID 38419787
- [Derived] Balasubramanian P, Kernan WN, Sheth KN, Ofstad AP, Rosenstock J, Wanner C, Zinman B, Mattheus M, Marx N, Inzucchi SE. Baseline Cardiovascular Risk Factor Control in Patients With Type 2 Diabetes and Coronary Disease Versus Stroke: Secondary Analysis of Cardiovascular Outcome Trials. Stroke. 2023 Aug;54(8):2013-2021. doi: 10.1161/STROKEAHA.122.042053. Epub 2023 Jul 14. PMID 37449424
- [Derived] Dar MS, Wanner C, Marx N, Ofstad AP, Mattheus M, Kaspers S, Beg SA. Cardiovascular outcomes trial data from EMPA-REG OUTCOME, CAROLINA and CARMELINA: Assessment of a novel staging system for type 2 diabetes. Diabetes Obes Metab. 2023 May;25(5):1372-1384. doi: 10.1111/dom.14989. Epub 2023 Mar 6. PMID 36700391
- [Derived] Tuttle KR, Levin A, Nangaku M, Kadowaki T, Agarwal R, Hauske SJ, Elsasser A, Ritter I, Steubl D, Wanner C, Wheeler DC. Safety of Empagliflozin in Patients With Type 2 Diabetes and Chronic Kidney Disease: Pooled Analysis of Placebo-Controlled Clinical Trials. Diabetes Care. 2022 Jun 2;45(6):1445-1452. doi: 10.2337/dc21-2034. PMID 35472672
- [Derived] Kahl S, Ofstad AP, Zinman B, Wanner C, Schuler E, Sattar N, Inzucchi SE, Roden M. Effects of empagliflozin on markers of liver steatosis and fibrosis and their relationship to cardiorenal outcomes. Diabetes Obes Metab. 2022 Jun;24(6):1061-1071. doi: 10.1111/dom.14670. Epub 2022 Mar 8. PMID 35166009
- [Derived] Ruggenenti P, Kraus BJ, Inzucchi SE, Zinman B, Hantel S, Mattheus M, von Eynatten M, Remuzzi G, Koitka-Weber A, Wanner C. Nephrotic-range proteinuria in type 2 diabetes: Effects of empagliflozin on kidney disease progression and clinical outcomes. EClinicalMedicine. 2021 Dec 24;43:101240. doi: 10.1016/j.eclinm.2021.101240. eCollection 2022 Jan. PMID 35005582
- [Derived] Reifsnider OS, Kansal AR, Wanner C, Pfarr E, Koitka-Weber A, Brand SB, Stargardter M, Wang C, Kuti E, Ustyugova A. Cost-Effectiveness of Empagliflozin in Patients With Diabetic Kidney Disease in the United States: Findings Based on the EMPA-REG OUTCOME Trial. Am J Kidney Dis. 2022 Jun;79(6):796-806. doi: 10.1053/j.ajkd.2021.09.014. Epub 2021 Nov 6. PMID 34752913
- [Derived] Ferreira JP, Inzucchi SE, Mattheus M, Meinicke T, Steubl D, Wanner C, Zinman B. Empagliflozin and uric acid metabolism in diabetes: A post hoc analysis of the EMPA-REG OUTCOME trial. Diabetes Obes Metab. 2022 Jan;24(1):135-141. doi: 10.1111/dom.14559. Epub 2021 Oct 4. PMID 34558768
- [Derived] Vaduganathan M, Inzucchi SE, Sattar N, Fitchett DH, Ofstad AP, Brueckmann M, George JT, Verma S, Mattheus M, Wanner C, Zinman B, Butler J. Effects of empagliflozin on insulin initiation or intensification in patients with type 2 diabetes and cardiovascular disease: Findings from the EMPA-REG OUTCOME trial. Diabetes Obes Metab. 2021 Dec;23(12):2775-2784. doi: 10.1111/dom.14535. Epub 2021 Oct 7. PMID 34463409
- [Derived] Sharma A, Ofstad AP, Ahmad T, Zinman B, Zwiener I, Fitchett D, Wanner C, George JT, Hantel S, Desai N, Mentz RJ. Patient Phenotypes and SGLT-2 Inhibition in Type 2 Diabetes: Insights From the EMPA-REG OUTCOME Trial. JACC Heart Fail. 2021 Aug;9(8):568-577. doi: 10.1016/j.jchf.2021.03.003. PMID 34325887
- [Derived] Cherney DZI, Dagogo-Jack S, McGuire DK, Cosentino F, Pratley R, Shih WJ, Frederich R, Maldonado M, Liu J, Wang S, Cannon CP; VERTIS CV Investigators. Kidney outcomes using a sustained >/=40% decline in eGFR: A meta-analysis of SGLT2 inhibitor trials. Clin Cardiol. 2021 Aug;44(8):1139-1143. doi: 10.1002/clc.23665. Epub 2021 Jun 15. PMID 34129237
- [Derived] Ferreira JP, Kraus BJ, Zwiener I, Lauer S, Zinman B, Fitchett DH, Koitka-Weber A, George JT, Ofstad AP, Wanner C, Zannad F. Cardio/Kidney Composite End Points: A Post Hoc Analysis of the EMPA-REG OUTCOME Trial. J Am Heart Assoc. 2021 Apr 6;10(7):e020053. doi: 10.1161/JAHA.120.020053. Epub 2021 Mar 23. PMID 33754809
- [Derived] Ferreira JP, Verma S, Fitchett D, Ofstad AP, Lauer S, Zwiener I, George J, Wanner C, Zinman B, Inzucchi SE. Metabolic syndrome in patients with type 2 diabetes and atherosclerotic cardiovascular disease: a post hoc analyses of the EMPA-REG OUTCOME trial. Cardiovasc Diabetol. 2020 Nov 26;19(1):200. doi: 10.1186/s12933-020-01174-6. PMID 33243221
- [Derived] McGuire DK, Zinman B, Inzucchi SE, Wanner C, Fitchett D, Anker SD, Pocock S, Kaspers S, George JT, von Eynatten M, Johansen OE, Jamal W, Mattheus M, Elsasser U, Hantel S, Lund SS. Effects of empagliflozin on first and recurrent clinical events in patients with type 2 diabetes and atherosclerotic cardiovascular disease: a secondary analysis of the EMPA-REG OUTCOME trial. Lancet Diabetes Endocrinol. 2020 Dec;8(12):949-959. doi: 10.1016/S2213-8587(20)30344-2. PMID 33217335
- [Derived] Ceriello A, Ofstad AP, Zwiener I, Kaspers S, George J, Nicolucci A. Empagliflozin reduced long-term HbA1c variability and cardiovascular death: insights from the EMPA-REG OUTCOME trial. Cardiovasc Diabetol. 2020 Oct 13;19(1):176. doi: 10.1186/s12933-020-01147-9. PMID 33050931
- [Derived] Neeland IJ, Eliasson B, Kasai T, Marx N, Zinman B, Inzucchi SE, Wanner C, Zwiener I, Wojeck BS, Yaggi HK, Johansen OE; EMPA-REG OUTCOME Investigators. The Impact of Empagliflozin on Obstructive Sleep Apnea and Cardiovascular and Renal Outcomes: An Exploratory Analysis of the EMPA-REG OUTCOME Trial. Diabetes Care. 2020 Dec;43(12):3007-3015. doi: 10.2337/dc20-1096. Epub 2020 Oct 1. PMID 33004464
- [Derived] Levin A, Perkovic V, Wheeler DC, Hantel S, George JT, von Eynatten M, Koitka-Weber A, Wanner C; EMPA-REG OUTCOME Investigators. Empagliflozin and Cardiovascular and Kidney Outcomes across KDIGO Risk Categories: Post Hoc Analysis of a Randomized, Double-Blind, Placebo-Controlled, Multinational Trial. Clin J Am Soc Nephrol. 2020 Oct 7;15(10):1433-1444. doi: 10.2215/CJN.14901219. Epub 2020 Sep 29. PMID 32994159
- [Derived] Waijer SW, Xie D, Inzucchi SE, Zinman B, Koitka-Weber A, Mattheus M, von Eynatten M, Inker LA, Wanner C, Heerspink HJL. Short-Term Changes in Albuminuria and Risk of Cardiovascular and Renal Outcomes in Type 2 Diabetes Mellitus: A Post Hoc Analysis of the EMPA-REG OUTCOME Trial. J Am Heart Assoc. 2020 Sep 15;9(18):e016976. doi: 10.1161/JAHA.120.016976. Epub 2020 Sep 6. PMID 32893717
- [Derived] Bohm M, Fitchett D, Ofstad AP, Brueckmann M, Kaspers S, George JT, Zwiener I, Zinman B, Wanner C, Marx N, Mancia G, Anker SD, Mahfoud F. Heart failure and renal outcomes according to baseline and achieved blood pressure in patients with type 2 diabetes: results from EMPA-REG OUTCOME. J Hypertens. 2020 Sep;38(9):1829-1840. doi: 10.1097/HJH.0000000000002492. PMID 32618884
- [Derived] Inzucchi SE, Khunti K, Fitchett DH, Wanner C, Mattheus M, George JT, Ofstad AP, Zinman B. Cardiovascular Benefit of Empagliflozin Across the Spectrum of Cardiovascular Risk Factor Control in the EMPA-REG OUTCOME Trial. J Clin Endocrinol Metab. 2020 Sep 1;105(9):3025-35. doi: 10.1210/clinem/dgaa321. PMID 32485734
- [Derived] Ferreira JP, Fitchett D, Ofstad AP, Kraus BJ, Wanner C, Zwiener I, Zinman B, Lauer S, George JT, Rossignol P, Zannad F. Empagliflozin for Patients With Presumed Resistant Hypertension: A Post Hoc Analysis of the EMPA-REG OUTCOME Trial. Am J Hypertens. 2020 Dec 31;33(12):1092-1101. doi: 10.1093/ajh/hpaa073. PMID 32369546
- [Derived] Perkovic V, Koitka-Weber A, Cooper ME, Schernthaner G, Pfarr E, Woerle HJ, von Eynatten M, Wanner C. Choice of endpoint in kidney outcome trials: considerations from the EMPA-REG OUTCOME(R) trial. Nephrol Dial Transplant. 2020 Dec 4;35(12):2103-2111. doi: 10.1093/ndt/gfz179. PMID 31495881
- [Derived] Kansal A, Reifsnider OS, Proskorovsky I, Zheng Y, Pfarr E, George JT, Kandaswamy P, Ruffolo A. Cost-effectiveness analysis of empagliflozin treatment in people with Type 2 diabetes and established cardiovascular disease in the EMPA-REG OUTCOME trial. Diabet Med. 2019 Nov;36(11):1494-1502. doi: 10.1111/dme.14076. Epub 2019 Jul 23. PMID 31295358
- [Derived] Butler J, Zannad F, Fitchett D, Zinman B, Koitka-Weber A, von Eynatten M, Zwiener I, George J, Brueckmann M, Cheung AK, Wanner C. Empagliflozin Improves Kidney Outcomes in Patients With or Without Heart Failure. Circ Heart Fail. 2019 Jun;12(6):e005875. doi: 10.1161/CIRCHEARTFAILURE.118.005875. Epub 2019 Jun 5. PMID 31163986
- [Derived] Verma S, Wanner C, Zwiener I, Ofstad AP, George JT, Fitchett D, Zinman B; EMPA-REG OUTCOME Investigators. Influence of Microvascular Disease on Cardiovascular Events in Type 2 Diabetes. J Am Coll Cardiol. 2019 Jun 4;73(21):2780-2782. doi: 10.1016/j.jacc.2019.03.002. Epub 2019 Mar 15. No abstract available. PMID 30885684
- [Derived] Januzzi J, Ferreira JP, Bohm M, Kaul S, Wanner C, Brueckmann M, Petrie MC, Ofstad AP, Zeller C, George J, Fitchett D, Zannad F. Empagliflozin reduces the risk of a broad spectrum of heart failure outcomes regardless of heart failure status at baseline. Eur J Heart Fail. 2019 Mar;21(3):386-388. doi: 10.1002/ejhf.1419. Epub 2019 Feb 14. No abstract available. PMID 30767353
- [Derived] Fitchett D, Inzucchi SE, Cannon CP, McGuire DK, Scirica BM, Johansen OE, Sambevski S, Kaspers S, Pfarr E, George JT, Zinman B. Empagliflozin Reduced Mortality and Hospitalization for Heart Failure Across the Spectrum of Cardiovascular Risk in the EMPA-REG OUTCOME Trial. Circulation. 2019 Mar 12;139(11):1384-1395. doi: 10.1161/CIRCULATIONAHA.118.037778. PMID 30586757
- [Derived] Verma S, Mazer CD, Fitchett D, Inzucchi SE, Pfarr E, George JT, Zinman B. Empagliflozin reduces cardiovascular events, mortality and renal events in participants with type 2 diabetes after coronary artery bypass graft surgery: subanalysis of the EMPA-REG OUTCOME(R) randomised trial. Diabetologia. 2018 Aug;61(8):1712-1723. doi: 10.1007/s00125-018-4644-9. Epub 2018 May 19. PMID 29777264
- [Derived] Wittbrodt ET, Eudicone JM, Bell KF, Enhoffer DM, Latham K, Green JB. Eligibility varies among the 4 sodium-glucose cotransporter-2 inhibitor cardiovascular outcomes trials: implications for the general type 2 diabetes US population. Am J Manag Care. 2018 Apr;24(8 Suppl):S138-S145. PMID 29693360
- [Derived] Inzucchi SE, Zinman B, Fitchett D, Wanner C, Ferrannini E, Schumacher M, Schmoor C, Ohneberg K, Johansen OE, George JT, Hantel S, Bluhmki E, Lachin JM. How Does Empagliflozin Reduce Cardiovascular Mortality? Insights From a Mediation Analysis of the EMPA-REG OUTCOME Trial. Diabetes Care. 2018 Feb;41(2):356-363. doi: 10.2337/dc17-1096. Epub 2017 Dec 4. PMID 29203583
- [Derived] Wanner C, Lachin JM, Inzucchi SE, Fitchett D, Mattheus M, George J, Woerle HJ, Broedl UC, von Eynatten M, Zinman B; EMPA-REG OUTCOME Investigators. Empagliflozin and Clinical Outcomes in Patients With Type 2 Diabetes Mellitus, Established Cardiovascular Disease, and Chronic Kidney Disease. Circulation. 2018 Jan 9;137(2):119-129. doi: 10.1161/CIRCULATIONAHA.117.028268. Epub 2017 Sep 13. PMID 28904068
- [Derived] Cherney DZI, Zinman B, Inzucchi SE, Koitka-Weber A, Mattheus M, von Eynatten M, Wanner C. Effects of empagliflozin on the urinary albumin-to-creatinine ratio in patients with type 2 diabetes and established cardiovascular disease: an exploratory analysis from the EMPA-REG OUTCOME randomised, placebo-controlled trial. Lancet Diabetes Endocrinol. 2017 Aug;5(8):610-621. doi: 10.1016/S2213-8587(17)30182-1. Epub 2017 Jun 27. PMID 28666775
- [Derived] Zinman B, Inzucchi SE, Lachin JM, Wanner C, Fitchett D, Kohler S, Mattheus M, Woerle HJ, Broedl UC, Johansen OE, Albers GW, Diener HC; EMPA-REG OUTCOME Investigators (Empagliflozin Cardiovascular Outcome Event Trial in Type 2 Diabetes Mellitus Patients). Empagliflozin and Cerebrovascular Events in Patients With Type 2 Diabetes Mellitus at High Cardiovascular Risk. Stroke. 2017 May;48(5):1218-1225. doi: 10.1161/STROKEAHA.116.015756. Epub 2017 Apr 6. PMID 28386035
- [Derived] Wanner C, Inzucchi SE, Lachin JM, Fitchett D, von Eynatten M, Mattheus M, Johansen OE, Woerle HJ, Broedl UC, Zinman B; EMPA-REG OUTCOME Investigators. Empagliflozin and Progression of Kidney Disease in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):323-34. doi: 10.1056/NEJMoa1515920. Epub 2016 Jun 14. PMID 27299675
- [Derived] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Derived] Zinman B, Inzucchi SE, Lachin JM, Wanner C, Ferrari R, Fitchett D, Bluhmki E, Hantel S, Kempthorne-Rawson J, Newman J, Johansen OE, Woerle HJ, Broedl UC. Rationale, design, and baseline characteristics of a randomized, placebo-controlled cardiovascular outcome trial of empagliflozin (EMPA-REG OUTCOME). Cardiovasc Diabetol. 2014 Jun 19;13:102. doi: 10.1186/1475-2840-13-102. PMID 24943000

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients randomised to treatments in 1:1:1 ratio.
Pre-assignment Details: Randomisation stratified by:BMI at randomisation(<30/≥30 kg/m2),HbA1c at screening (<8.5%/ ≥8.5%);geographical region(North America including Australia and New Zealand,Latin America,Europe,Africa,Asia);renal function at screening (normal:eGFR ≥90 mL/min, mild impairment:60 mL/min ≤ eGFR ≤89 mL/min, moderate impairment:30 mL/min ≤ eGFR≤59 mL/min).
Groups:
- Placebo: Oral administration of Placebo matching empagliflozin 10 mg or 25 mg (1 tablet once daily)
- Empagliflozin 10 mg: Oral administration of Empagliflozin 10 mg (BI 10773) film coated tablets (1 tablet once daily)
- Empagliflozin 25 mg: Oral administration of Empagliflozin 25 mg (BI 10773) film coated tablets (1 tablet once daily)
Period: Discontinuation From Treatment
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Started | 2337 (Randomised) | 2347 (Randomised) | 2344 (Randomised)
Completed | 1650 (Not prematurely discontinued from trial medication) | 1790 (Not prematurely discontinued from trial medication) | 1800 (Not prematurely discontinued from trial medication)
Not Completed | 687 | 557 | 544
Not completed — Study drug stopped, reason missing | 5 | 3 | 4
Not completed — Not treated | 4 | 2 | 2
Not completed — Lack of Efficacy | 11 | 1 | 0
Not completed — Non compliant with protocol | 15 | 15 | 12
Not completed — Lost to Follow-up | 15 | 9 | 6
Not completed — Refusal to continue, not due to AE | 172 | 118 | 122
Not completed — Other than those specified | 162 | 142 | 125
Not completed — Adverse Event | 303 | 267 | 273
Period: Discontinuation From Study (Treated Set)
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Started | 2333 | 2345 | 2342
Final Vital Status (VS) Available | 2316 | 2324 | 2327
Completed | 2266 (Completed the trial or died) | 2264 (Completed the trial or died) | 2279 (Completed the trial or died)
Not Completed | 67 | 81 | 63
Not completed — Consent withdrawn: Final VS available | 23 | 35 | 25
Not completed — Consent withdrawn:Final VS not available | 8 | 6 | 5
Not completed — Site closure: Final VS available | 20 | 21 | 19
Not completed — Site closure:Final VS not available (NA) | 5 | 9 | 7
Not completed — Lost to FU for 3PMACE:Final VS available | 7 | 6 | 5
Not completed — Lost to FU for 3P-MACE:Final VS NA | 4 | 4 | 2

BASELINE CHARACTERISTICS:
Population: Treated set (TS): Consists of all randomised patients who received at least 1 dose of study medication. Patients were assigned to treatment groups according to the randomisation scheme.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg | Total
Number analyzed (Participants) | 2333 | 2345 | 2342 | 7020
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (8.8) | 63.0 (8.6) | 63.2 (8.6) | 63.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 653 | 692 | 659 | 2004
  Male | 1680 | 1653 | 1683 | 5016

OUTCOME MEASURES:

1. Primary Outcome: Time to the First Occurrence of Any of the Following Adjudicated Components of the Primary Composite Endpoint (3-point MACE): CV Death (Including Fatal Stroke and Fatal MI), Non-fatal MI (Excluding Silent MI), and Non-fatal Stroke.
Description: Time to the first occurrence of any of the following adjudicated components of the primary composite endpoint (3-point major adverse cardiovascular events (MACE)): cardiovascular (CV) death (including fatal stroke and fatal myocardial infarction (MI)), non-fatal MI (excluding silent MI), and non-fatal stroke.
  Percentage of patients with the event are presented.
Time Frame: From randomisation to individual end of observation, up to 4.6 years
Population: TS
Measure: Number; unit: percentage of participants
Groups:
- All Empagliflozin: Patients who received either 10 mg or 25 mg of empagliflozin were pooled into a common empagliflozin treatment group
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg | All Empagliflozin
Number analyzed (Participants) | 2333 | 2345 | 2342 | 4687
percentage of participants | 12.1 | 10.4 | 10.5 | 10.5
Statistical Analysis 1: Comparison: Placebo vs All Empagliflozin; Primary objective was to establish the non-inferiority of All empagliflozin relative to placebo for time to first 3-point MACE. A 4-step hierarchical testing strategy was followed for the non-inferiority test of the primary endpoint and then the key secondary endpoint, each at a margin of 1.3, followed by test of superiority of primary and key secondary endpoints; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was chosen as 1.3 based on Food and Drug Administration (FDA) Guidance for Industry - Diabetes Mellitus - Evaluating Cardiovascular Risk in New Antidiabetic Therapies to Treat Type 2 Diabetes; p < 0.0001, Cox proportional hazards model — One-sided test with alpha = 0.0249; Cox proportional hazards model with factors for treatment, age, gender, categorised BMI, HbA1c, eGFR and geographical region; Hazard Ratio (HR) = 0.86, 95.02% CI 2-sided [0.74 to 0.99] — All Empagliflozin divided by Placebo
Statistical Analysis 2: Comparison: Placebo vs All Empagliflozin; Test type: Superiority or Other; p = 0.0382, Cox proportional hazards model — Two-sided test with alpha=0.0498; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.86, 95.02% CI 2-sided [0.74 to 0.99] — All Empagliflozin divided by Placebo

2. Secondary Outcome: Percentage of Participants With the Composite of All Events Adjudicated (4-point MACE): CV Death (Including Fatal Stroke and Fatal MI), Non-fatal MI (Excluding Silent MI), Non-fatal Stroke and Hospitalization for Unstable Angina Pectoris
Description: The composite of all events adjudicated (4-point MACE): cardiovascular death (including fatal stroke and fatal myocardial infarction), non-fatal myocardial infarction (excluding silent MI), non-fatal stroke and hospitalization for unstable angina pectoris.This is a key secondary endpoint of the trial.
  Percentage of patients with the event are presented.
Time Frame: From randomisation to individual end of observation, up to 4.6 years
Population: TS
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg | All Empagliflozin
Number analyzed (Participants) | 2333 | 2345 | 2342 | 4687
percentage of participants | 14.3 | 12.8 | 12.8 | 12.8
Statistical Analysis 1: Comparison: Placebo vs All Empagliflozin; A 4-step hierarchical testing strategy was followed for the non-inferiority test of the primary endpoint and then the key secondary endpoint, each at a margin of 1.3, followed by test of superiority of primary and key secondary endpoints; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cox proportional hazards model — One-sided test with alpha = 0.0249; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.89, 95.02% CI 2-sided [0.78 to 1.01] — All Empagliflozin divided by Placebo
Statistical Analysis 2: Comparison: Placebo vs All Empagliflozin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0795, Cox proportional hazards model — Two-sided test with alpha=0.0498; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.89, 95.02% CI 2-sided [0.78 to 1.01] — All Empagliflozin divided by Placebo

3. Secondary Outcome: Percentage of Participants With Silent MI
Description: Silent MI; defined as presence in the ECG of:
  * Any Q-wave in leads V2-V3 ≥0.02 seconds or QS complex in leads V2 and V3
  * Q-wave ≥0.03 seconds and ≥0.1 mV deep or QS complex in leads I, II, aVL, aVF, or V4-V6 in any two leads of a contiguous lead grouping (I, aVL, V6; V4-V6; II, III, and aVF)
  * R-wave ≥0.04 seconds in V1-V2 and R/S ≥1 with a concordant positive T-wave in the absence of a conduction defect.
  It was also required that there had been no adjudicated and confirmed event of either acute MI, hospitalisation for unstable angina, coronary revascularisation procedures or stent thrombosis following randomisation up to and including the date of the specified ECG measurement.
  Percentage of patients with the event are presented.
Time Frame: From randomisation to individual end of observation, up to 4.6 years
Population: TS (evaluable cases)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg | All Empagliflozin
Number analyzed (Participants) | 1211 | 1174 | 1204 | 2378
percentage of participants | 1.2 | 1.6 | 1.6 | 1.6
Statistical Analysis 1: Comparison: Placebo vs All Empagliflozin; Test type: Superiority or Other; p = 0.4172, Cox proportional hazards model — Two-sided test with alpha = 0.05; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.28, 95% CI 2-sided [0.70 to 2.33] — All Empagliflozin divided by Placebo

4. Secondary Outcome: Percentage of Participants With Heart Failure Requiring Hospitalisation (Adjudicated)
Description: Heart failure requiring hospitalisation (adjudicated). Percentage of patients with the event are presented.
Time Frame: From randomisation to individual end of observation, up to 4.6 years
Population: TS
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg | All Empagliflozin
Number analyzed (Participants) | 2333 | 2345 | 2342 | 4687
percentage of participants | 4.1 | 2.6 | 2.8 | 2.7
Statistical Analysis 1: Comparison: Placebo vs All Empagliflozin; Test type: Superiority or Other; p = 0.0017, Cox proportional hazards model — Two-sided test with alpha = 0.05; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.50 to 0.85] — All Empagliflozin divided by Placebo

5. Secondary Outcome: Percentage of Participants With New Onset Albuminuria
Description: New onset albuminuria defined as urine albumin / creatinine ratio (UACR) ≥30 mg/g.
  Percentage of patients with the event are presented.
Time Frame: From randomisation to individual end of observation, up to 4.6 years
Population: TS (evaluable cases)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg | All Empagliflozin
Number analyzed (Participants) | 1374 | 1403 | 1376 | 2779
percentage of participants | 51.2 | 51.5 | 51.5 | 51.5
Statistical Analysis 1: Comparison: Placebo vs All Empagliflozin; Test type: Superiority or Other; p = 0.2547, Cox proportional hazards model — Two-sided test with alpha = 0.05; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.87 to 1.04] — All Empagliflozin divided by Placebo

6. Secondary Outcome: Percentage of Participants With New Onset Macroalbuminuria
Description: New onset macroalbuminuria defined as UACR >300 mg/g. Percentage of patients with the event are presented.
Time Frame: From randomisation to individual end of observation, up to 4.6 years
Population: TS (evaluable cases)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg | All Empagliflozin
Number analyzed (Participants) | 2033 | 2037 | 2054 | 4091
percentage of participants | 16.2 | 10.9 | 11.5 | 11.2
Statistical Analysis 1: Comparison: Placebo vs All Empagliflozin; Test type: Superiority or Other; p < 0.0001, Cox proportional hazards model — Two-sided test with alpha = 0.05; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.54 to 0.72] — All Empagliflozin divided by Placebo

7. Secondary Outcome: Percentage of Participants With the Composite Microvascular Outcome
Description: Composite microvascular outcome defined as:
  * Initiation of retinal photocoagulation
  * Vitreous haemorrhage
  * Diabetes-related blindness, or
  * New or worsening nephropathy defined as:
    * New onset of macroalbuminuria; or
    * Doubling of serum creatinine level accompanied by an eGFR (based on modification of diet in renal disease (MDRD) formula) ≤45 mL/min/1.73m2; or
    * Initiation of continuous renal replacement therapy, or
    * Death due to renal disease. Percentage of patients with the event are presented.
Time Frame: From randomisation to individual end of observation, up to 4.6 years
Population: TS (evaluable cases)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg | All Empagliflozin
Number analyzed (Participants) | 2068 | 2057 | 2075 | 4132
percentage of participants | 20.5 | 13.9 | 14.1 | 14.0
Statistical Analysis 1: Comparison: Placebo vs All Empagliflozin; Test type: Superiority or Other; p < 0.0001, Cox proportional hazards model — Two-sided test with alpha = 0.05; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.54 to 0.70] — All Empagliflozin divided by Placebo

ADVERSE EVENTS:
Time Frame: All AEs, serious and non-serious, occurring during the course of the clinical trial (from randomisation through the follow-up period); up to 5 years
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Serious Adverse Events (participants affected / at risk) | 988/2333 | 876/2345 | 913/2342
Other Adverse Events (participants affected / at risk) | 1690/2333 | 1556/2345 | 1551/2342
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=2333) | Empagliflozin 10 mg (N=2345) | Empagliflozin 25 mg (N=2342)
Anaemia (Blood and lymphatic system disorders) | 12 | 8 | 7
Coagulopathy (Blood and lymphatic system disorders) | 1 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Hypereosinophilic syndrome (Blood and lymphatic system disorders) | 1 | 0 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Hypocoagulable state (Blood and lymphatic system disorders) | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 1 | 4
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 10 | 10 | 14
Acute myocardial infarction (Cardiac disorders) | 42 | 32 | 48
Angina pectoris (Cardiac disorders) | 32 | 36 | 42
Angina unstable (Cardiac disorders) | 87 | 82 | 73
Aortic valve disease (Cardiac disorders) | 0 | 0 | 2
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 2
Arrhythmia (Cardiac disorders) | 2 | 5 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 1 | 6
Atrial fibrillation (Cardiac disorders) | 14 | 25 | 12
Atrial flutter (Cardiac disorders) | 5 | 7 | 4
Atrial tachycardia (Cardiac disorders) | 1 | 1 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block (Cardiac disorders) | 3 | 2 | 1
Atrioventricular block complete (Cardiac disorders) | 2 | 2 | 3
Atrioventricular block first degree (Cardiac disorders) | 1 | 1 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 2 | 1
Bradyarrhythmia (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 11 | 2 | 4
Bundle branch block bilateral (Cardiac disorders) | 0 | 0 | 1
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 12 | 6 | 5
Cardiac asthma (Cardiac disorders) | 0 | 1 | 0
Cardiac disorder (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 55 | 42 | 24
Cardiac failure acute (Cardiac disorders) | 9 | 4 | 2
Cardiac failure chronic (Cardiac disorders) | 0 | 4 | 2
Cardiac failure congestive (Cardiac disorders) | 45 | 30 | 35
Cardiac failure high output (Cardiac disorders) | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 6 | 5 | 2
Cardiogenic shock (Cardiac disorders) | 2 | 2 | 2
Cardiomyopathy (Cardiac disorders) | 2 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 2 | 0 | 1
Cardiorenal syndrome (Cardiac disorders) | 0 | 0 | 1
Cardiovascular disorder (Cardiac disorders) | 1 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 46 | 21 | 29
Coronary artery insufficiency (Cardiac disorders) | 1 | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 6 | 3 | 7
Coronary artery stenosis (Cardiac disorders) | 5 | 5 | 5
Cyanosis (Cardiac disorders) | 1 | 0 | 0
Diastolic dysfunction (Cardiac disorders) | 2 | 0 | 0
Hypertensive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 1 | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0 | 4
Left atrial dilatation (Cardiac disorders) | 0 | 1 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 2
Left ventricular failure (Cardiac disorders) | 2 | 1 | 0
Microvascular coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 47 | 50 | 44
Myocardial ischaemia (Cardiac disorders) | 15 | 5 | 7
Myocarditis (Cardiac disorders) | 1 | 0 | 0
Nodal arrhythmia (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 2 | 1
Papillary muscle disorder (Cardiac disorders) | 1 | 0 | 0
Pericardial cyst (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 2 | 2 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Postinfarction angina (Cardiac disorders) | 1 | 0 | 1
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0
Silent myocardial infarction (Cardiac disorders) | 1 | 3 | 3
Sinus arrhythmia (Cardiac disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 1 | 2
Sinus node dysfunction (Cardiac disorders) | 6 | 5 | 3
Supraventricular tachycardia (Cardiac disorders) | 4 | 5 | 1
Systolic dysfunction (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 5 | 3 | 0
Tachycardia paroxysmal (Cardiac disorders) | 1 | 0 | 0
Trifascicular block (Cardiac disorders) | 1 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 2 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 2 | 1 | 2
Ventricular tachycardia (Cardiac disorders) | 8 | 2 | 5
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 0
Congenital anomalies of ear ossicles (Congenital, familial and genetic disorders) | 1 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 1 | 1 | 2
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 7 | 2 | 9
Vertigo positional (Ear and labyrinth disorders) | 6 | 0 | 2
Basedow's disease (Endocrine disorders) | 0 | 1 | 0
Goitre (Endocrine disorders) | 1 | 0 | 2
Hyperparathyroidism (Endocrine disorders) | 0 | 1 | 2
Hyperparathyroidism primary (Endocrine disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Amaurosis (Eye disorders) | 0 | 1 | 0
Blindness (Eye disorders) | 1 | 0 | 0
Blindness unilateral (Eye disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 9 | 13 | 11
Cataract cortical (Eye disorders) | 1 | 0 | 0
Corneal degeneration (Eye disorders) | 0 | 0 | 1
Diabetic retinopathy (Eye disorders) | 4 | 1 | 2
Exfoliation syndrome (Eye disorders) | 0 | 0 | 1
Glaucoma (Eye disorders) | 1 | 3 | 2
Keratopathy (Eye disorders) | 0 | 0 | 1
Macular fibrosis (Eye disorders) | 1 | 0 | 0
Macular oedema (Eye disorders) | 2 | 1 | 0
Papilloedema (Eye disorders) | 1 | 0 | 0
Retinal artery occlusion (Eye disorders) | 0 | 1 | 2
Retinal detachment (Eye disorders) | 0 | 4 | 2
Retinal haemorrhage (Eye disorders) | 1 | 0 | 0
Retinal tear (Eye disorders) | 0 | 0 | 1
Retinopathy (Eye disorders) | 1 | 0 | 0
Retinoschisis (Eye disorders) | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 4 | 1 | 3
Vitreous opacities (Eye disorders) | 0 | 3 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 2 | 2
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 5 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3 | 2
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 2 | 0
Bezoar (Gastrointestinal disorders) | 0 | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 2 | 3
Colitis ischaemic (Gastrointestinal disorders) | 1 | 1 | 0
Colon dysplasia (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 4 | 2 | 2
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 0 | 1
Diabetic gastropathy (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 6 | 4
Diverticulum (Gastrointestinal disorders) | 2 | 1 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 3 | 1
Duodenal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 2 | 2 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Erosive duodenitis (Gastrointestinal disorders) | 1 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 2 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 2
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 3 | 1 | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 2 | 7
Gastritis erosive (Gastrointestinal disorders) | 1 | 1 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 9 | 4 | 4
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 7 | 3
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 2 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 3 | 2 | 1
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 1
Ileus paralytic (Gastrointestinal disorders) | 3 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 3
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 3 | 5 | 4
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 | 1 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 2 | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 5 | 1 | 3
Intestinal perforation (Gastrointestinal disorders) | 2 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 5 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 | 1 | 0
Lumbar hernia (Gastrointestinal disorders) | 0 | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 1 | 1
Melaena (Gastrointestinal disorders) | 0 | 1 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 4 | 2
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 4 | 3 | 3
Pancreatitis acute (Gastrointestinal disorders) | 3 | 1 | 3
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis relapsing (Gastrointestinal disorders) | 1 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 2 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Peptic ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 3 | 2
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Stress ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 2 | 3 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 2 | 5
Varices oesophageal (Gastrointestinal disorders) | 0 | 1 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3 | 4
Adverse drug reaction (General disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 2 | 1
Cardiac death (General disorders) | 3 | 4 | 2
Chest discomfort (General disorders) | 4 | 2 | 3
Chest pain (General disorders) | 28 | 32 | 33
Chills (General disorders) | 1 | 0 | 0
Death (General disorders) | 12 | 10 | 5
Device defective (General disorders) | 1 | 0 | 0
Device deposit issue (General disorders) | 1 | 0 | 0
Device difficult to use (General disorders) | 1 | 0 | 0
Device malfunction (General disorders) | 1 | 0 | 0
Device occlusion (General disorders) | 0 | 0 | 2
Drowning (General disorders) | 0 | 1 | 0
Drug ineffective (General disorders) | 0 | 0 | 1
Dysplasia (General disorders) | 0 | 1 | 0
Extravasation (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0
Feeling abnormal (General disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 1 | 1 | 1
General physical health deterioration (General disorders) | 2 | 0 | 1
Generalised oedema (General disorders) | 1 | 0 | 0
Granuloma (General disorders) | 1 | 0 | 0
Hernia (General disorders) | 2 | 0 | 0
Impaired healing (General disorders) | 0 | 1 | 1
Implant site necrosis (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 1
Multi-organ failure (General disorders) | 3 | 2 | 0
Necrobiosis (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 6 | 5 | 15
Oedema peripheral (General disorders) | 5 | 1 | 1
Oversensing (General disorders) | 2 | 0 | 0
Pacemaker generated arrhythmia (General disorders) | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0
Perforated ulcer (General disorders) | 1 | 0 | 1
Peripheral swelling (General disorders) | 2 | 1 | 1
Polyp (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 5 | 7 | 2
Stent malfunction (General disorders) | 0 | 0 | 1
Strangulated hernia (General disorders) | 0 | 0 | 1
Sudden cardiac death (General disorders) | 2 | 2 | 2
Sudden death (General disorders) | 6 | 8 | 5
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0
Ulcer (General disorders) | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 4 | 2
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 4 | 4 | 5
Cholecystitis acute (Hepatobiliary disorders) | 4 | 7 | 6
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 7 | 9 | 12
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 2 | 2 | 2
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | 0
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Portal hypertension (Hepatobiliary disorders) | 0 | 1 | 0
Post cholecystectomy syndrome (Hepatobiliary disorders) | 1 | 0 | 0
Sphincter of Oddi dysfunction (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1 | 1
Contrast media allergy (Immune system disorders) | 1 | 0 | 0
Food allergy (Immune system disorders) | 1 | 0 | 2
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Iodine allergy (Immune system disorders) | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 2 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 2 | 1
Abscess (Infections and infestations) | 0 | 1 | 0
Abscess limb (Infections and infestations) | 3 | 6 | 2
Abscess of eyelid (Infections and infestations) | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 2
Amoebiasis (Infections and infestations) | 0 | 1 | 0
Amoebic dysentery (Infections and infestations) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 1
Appendicitis (Infections and infestations) | 3 | 5 | 3
Appendicitis perforated (Infections and infestations) | 0 | 0 | 2
Arteriosclerotic gangrene (Infections and infestations) | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 1 | 2
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 2 | 0 | 3
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1
Biliary tract infection (Infections and infestations) | 1 | 0 | 0
Bone abscess (Infections and infestations) | 1 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 10 | 5 | 5
Bronchitis viral (Infections and infestations) | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 3 | 1 | 3
Catheter site infection (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 20 | 11 | 17
Cellulitis gangrenous (Infections and infestations) | 0 | 2 | 0
Cellulitis of male external genital organ (Infections and infestations) | 0 | 1 | 0
Cellulitis staphylococcal (Infections and infestations) | 0 | 1 | 0
Cholecystitis infective (Infections and infestations) | 0 | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 0 | 3
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 1
Cutaneous larva migrans (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 2 | 0 | 0
Cystitis bacterial (Infections and infestations) | 1 | 0 | 0
Dengue fever (Infections and infestations) | 1 | 2 | 1
Device related infection (Infections and infestations) | 1 | 0 | 0
Device related sepsis (Infections and infestations) | 1 | 0 | 0
Diabetic foot infection (Infections and infestations) | 6 | 5 | 7
Diabetic gangrene (Infections and infestations) | 3 | 1 | 2
Diverticulitis (Infections and infestations) | 3 | 3 | 0
Ear infection (Infections and infestations) | 1 | 0 | 1
Eczema infected (Infections and infestations) | 1 | 0 | 0
Empyema (Infections and infestations) | 1 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 1
Endophthalmitis (Infections and infestations) | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0
Enterocolitis viral (Infections and infestations) | 0 | 1 | 0
Epididymitis (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 9 | 8 | 5
Escherichia sepsis (Infections and infestations) | 2 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0
Febrile infection (Infections and infestations) | 0 | 0 | 1
Furuncle (Infections and infestations) | 1 | 0 | 0
Gallbladder empyema (Infections and infestations) | 1 | 0 | 0
Gangrene (Infections and infestations) | 8 | 10 | 6
Gastroenteritis (Infections and infestations) | 15 | 18 | 15
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Gastrointestinal protozoal infection (Infections and infestations) | 1 | 0 | 0
Giardiasis (Infections and infestations) | 0 | 0 | 1
H1N1 influenza (Infections and infestations) | 0 | 1 | 2
Incision site infection (Infections and infestations) | 0 | 0 | 1
Infected skin ulcer (Infections and infestations) | 4 | 2 | 3
Infectious colitis (Infections and infestations) | 0 | 0 | 1
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 2 | 0 | 0
Infusion site infection (Infections and infestations) | 0 | 1 | 0
Inguinal hernia gangrenous (Infections and infestations) | 0 | 0 | 1
Intestinal fistula infection (Infections and infestations) | 0 | 0 | 1
Intestinal tuberculosis (Infections and infestations) | 1 | 0 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0
Klebsiella infection (Infections and infestations) | 0 | 0 | 1
Labyrinthitis (Infections and infestations) | 1 | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 3 | 1 | 0
Localised infection (Infections and infestations) | 5 | 2 | 4
Lower respiratory tract infection (Infections and infestations) | 4 | 8 | 2
Lower respiratory tract infection bacterial (Infections and infestations) | 2 | 0 | 0
Lung infection (Infections and infestations) | 0 | 2 | 0
Lyme disease (Infections and infestations) | 0 | 0 | 1
Mediastinitis (Infections and infestations) | 2 | 0 | 1
Meningitis (Infections and infestations) | 1 | 0 | 0
Meningitis bacterial (Infections and infestations) | 0 | 1 | 0
Meningitis streptococcal (Infections and infestations) | 1 | 0 | 0
Meningitis tuberculous (Infections and infestations) | 1 | 0 | 0
Muscle abscess (Infections and infestations) | 0 | 0 | 1
Myelitis (Infections and infestations) | 0 | 1 | 0
Nasal abscess (Infections and infestations) | 0 | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 5 | 5 | 9
Osteomyelitis acute (Infections and infestations) | 0 | 0 | 1
Osteomyelitis bacterial (Infections and infestations) | 1 | 0 | 0
Osteomyelitis chronic (Infections and infestations) | 0 | 0 | 1
Otitis externa (Infections and infestations) | 1 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Periodontitis (Infections and infestations) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 2 | 3
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 1
Pertussis (Infections and infestations) | 1 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 53 | 41 | 38
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 1
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0
Pneumonia haemophilus (Infections and infestations) | 1 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 2 | 1 | 0
Post procedural sepsis (Infections and infestations) | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 1 | 2
Prostatic abscess (Infections and infestations) | 0 | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 1 | 0 | 0
Psoas abscess (Infections and infestations) | 1 | 0 | 0
Pulmonary mycosis (Infections and infestations) | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 2 | 1 | 0
Pyelonephritis (Infections and infestations) | 2 | 0 | 5
Pyelonephritis acute (Infections and infestations) | 6 | 4 | 1
Pyelonephritis chronic (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 7 | 0 | 2
Rhinitis (Infections and infestations) | 0 | 1 | 0
Rotavirus infection (Infections and infestations) | 0 | 1 | 0
Salmonellosis (Infections and infestations) | 2 | 0 | 0
Scrotal abscess (Infections and infestations) | 0 | 1 | 1
Sepsis (Infections and infestations) | 5 | 7 | 6
Septic encephalopathy (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 8 | 2 | 5
Sinusitis (Infections and infestations) | 1 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 2 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1
Staphylococcal skin infection (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 2
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 1 | 2 | 0
Tuberculosis (Infections and infestations) | 0 | 1 | 0
Tuberculous pleurisy (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 2
Urinary tract infection (Infections and infestations) | 16 | 13 | 16
Urinary tract infection fungal (Infections and infestations) | 0 | 0 | 3
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 3 | 6 | 11
Vaginal cellulitis (Infections and infestations) | 0 | 1 | 0
Varicella (Infections and infestations) | 1 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 2 | 0 | 1
Viral infection (Infections and infestations) | 0 | 2 | 5
Wound infection (Infections and infestations) | 3 | 4 | 3
Wound sepsis (Infections and infestations) | 0 | 0 | 1
Accident at work (Injury, poisoning and procedural complications) | 1 | 0 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 2 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 4 | 2
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 1 | 1
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Chemical poisoning (Injury, poisoning and procedural complications) | 1 | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 4 | 2 | 2
Coronary artery restenosis (Injury, poisoning and procedural complications) | 4 | 4 | 2
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 2
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 16 | 9 | 16
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 3 | 0 | 2
Fibula fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 0 | 1
Gastrointestinal anastomotic complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 2 | 1 | 7
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 2 | 3
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 2 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Kidney rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 3 | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Open fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Periorbital contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 1 | 2 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 3 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 3 | 0
Rib fracture (Injury, poisoning and procedural complications) | 6 | 4 | 4
Road traffic accident (Injury, poisoning and procedural complications) | 6 | 6 | 9
Scar (Injury, poisoning and procedural complications) | 0 | 1 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 3
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Stab wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 2 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 7 | 0 | 2
Tongue injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 | 2 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 2 | 0 | 0
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic renal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Vascular graft occlusion (Injury, poisoning and procedural complications) | 2 | 1 | 3
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 2
Wound (Injury, poisoning and procedural complications) | 2 | 3 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Angiogram (Investigations) | 1 | 0 | 1
Angiogram normal (Investigations) | 1 | 0 | 0
Anticoagulation drug level above therapeutic (Investigations) | 0 | 1 | 0
Arteriogram coronary (Investigations) | 2 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Biopsy lung (Investigations) | 1 | 0 | 1
Blood calcium decreased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase MB increased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 0
Blood creatinine increased (Investigations) | 2 | 1 | 2
Blood glucose fluctuation (Investigations) | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 1
Blood magnesium decreased (Investigations) | 1 | 0 | 0
Blood potassium increased (Investigations) | 2 | 0 | 1
Blood pressure increased (Investigations) | 2 | 0 | 0
Blood pressure orthostatic decreased (Investigations) | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 2 | 0
Cardiac murmur (Investigations) | 0 | 1 | 0
Cardiac stress test abnormal (Investigations) | 0 | 0 | 1
Catheterisation cardiac (Investigations) | 1 | 2 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 2 | 1 | 0
Heart rate irregular (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 3 | 0
Lipase increased (Investigations) | 2 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1
Oxygen consumption increased (Investigations) | 1 | 0 | 0
Physical examination (Investigations) | 0 | 0 | 1
Prostatic specific antigen increased (Investigations) | 0 | 0 | 1
Scan myocardial perfusion abnormal (Investigations) | 2 | 0 | 1
Smear cervix abnormal (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 1
Troponin I increased (Investigations) | 1 | 0 | 0
Troponin increased (Investigations) | 1 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 2
White blood cell count increased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 5 | 5 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 6 | 3 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 6 | 8 | 3
Diabetic complication (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 3 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 14 | 5 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 2 | 3
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 17 | 10 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Insulin resistance (Metabolism and nutrition disorders) | 1 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Lipomatosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 2
Obesity (Metabolism and nutrition disorders) | 3 | 2 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 3 | 8
Bone fistula (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dactylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Fracture delayed union (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Gouty tophus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 10 | 4 | 6
Lower extremity mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteitis deformans (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 15 | 15 | 17
Osteomalacia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 3 | 6
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 5
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 6 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 6 | 2 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 2
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 3
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 | 15 | 12
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Benign neoplasm of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign respiratory tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 5
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Bone giant cell tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 2
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 3
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Fibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Genital neoplasm malignant female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 1
Hodgkin's disease stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Large cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5 | 3
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 7
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 3
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5 | 5
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-Hodgkin's lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
POEMS syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Papillary serous endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 11 | 9
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 3
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1
Renal cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Splenic marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 6 | 3
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 4 | 3
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 1
Amnesia (Nervous system disorders) | 1 | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0
Autonomic neuropathy (Nervous system disorders) | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 1
Brain stem haemorrhage (Nervous system disorders) | 0 | 1 | 0
Brain stem infarction (Nervous system disorders) | 0 | 1 | 2
Brain stem ischaemia (Nervous system disorders) | 1 | 0 | 0
Brain stem stroke (Nervous system disorders) | 0 | 0 | 1
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0 | 0
Carotid artery disease (Nervous system disorders) | 0 | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 1 | 0 | 4
Carotid artery stenosis (Nervous system disorders) | 10 | 7 | 12
Carotid artery thrombosis (Nervous system disorders) | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 3 | 1 | 1
Central nervous system inflammation (Nervous system disorders) | 0 | 0 | 1
Cerebellar infarction (Nervous system disorders) | 1 | 2 | 2
Cerebral arteriosclerosis (Nervous system disorders) | 1 | 0 | 0
Cerebral artery occlusion (Nervous system disorders) | 1 | 1 | 1
Cerebral artery stenosis (Nervous system disorders) | 0 | 0 | 1
Cerebral ataxia (Nervous system disorders) | 1 | 0 | 1
Cerebral infarction (Nervous system disorders) | 7 | 7 | 11
Cerebral ischaemia (Nervous system disorders) | 1 | 3 | 1
Cerebrovascular accident (Nervous system disorders) | 31 | 46 | 37
Cerebrovascular disorder (Nervous system disorders) | 2 | 1 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1 | 0
Cervical cord compression (Nervous system disorders) | 1 | 0 | 0
Cervical myelopathy (Nervous system disorders) | 1 | 0 | 2
Cervical radiculopathy (Nervous system disorders) | 2 | 1 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 2
Complex partial seizures (Nervous system disorders) | 1 | 0 | 0
Coordination abnormal (Nervous system disorders) | 0 | 0 | 1
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 2 | 2 | 1
Dizziness (Nervous system disorders) | 5 | 8 | 5
Dysarthria (Nervous system disorders) | 0 | 1 | 0
Embolic cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Embolic stroke (Nervous system disorders) | 3 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 2 | 2
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 2 | 0 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 4 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 2
Hemiplegia (Nervous system disorders) | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0
Hypercapnic coma (Nervous system disorders) | 1 | 0 | 0
Hyperkinesia (Nervous system disorders) | 1 | 0 | 0
Hypertensive encephalopathy (Nervous system disorders) | 2 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 1
Hypoglycaemic coma (Nervous system disorders) | 0 | 0 | 1
Hypotonia (Nervous system disorders) | 0 | 1 | 0
IIIrd nerve paralysis (Nervous system disorders) | 0 | 0 | 1
Intercostal neuralgia (Nervous system disorders) | 1 | 0 | 2
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 22 | 18 | 20
Lacunar infarction (Nervous system disorders) | 2 | 1 | 2
Leukoencephalopathy (Nervous system disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 2 | 0 | 2
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 1
Mononeuritis (Nervous system disorders) | 1 | 0 | 0
Monoplegia (Nervous system disorders) | 1 | 0 | 0
Muscle spasticity (Nervous system disorders) | 0 | 1 | 0
Myelitis transverse (Nervous system disorders) | 0 | 0 | 1
Myelopathy (Nervous system disorders) | 0 | 0 | 1
Myoclonus (Nervous system disorders) | 0 | 1 | 1
Nerve root compression (Nervous system disorders) | 0 | 1 | 0
Neuroleptic malignant syndrome (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 1
Paraplegia (Nervous system disorders) | 0 | 1 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0 | 0
Partial seizures (Nervous system disorders) | 2 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 1 | 0 | 0
Petit mal epilepsy (Nervous system disorders) | 0 | 0 | 1
Piriformis syndrome (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 1
Radiculopathy (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 2 | 1
Seizure (Nervous system disorders) | 4 | 7 | 5
Sensory disturbance (Nervous system disorders) | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1
Spinal epidural haematoma (Nervous system disorders) | 0 | 0 | 1
Spondylitic myelopathy (Nervous system disorders) | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 3 | 3 | 2
Subdural hygroma (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 8 | 9 | 18
Thalamic infarction (Nervous system disorders) | 1 | 1 | 0
Thrombotic cerebral infarction (Nervous system disorders) | 1 | 0 | 1
Thrombotic stroke (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 23 | 23 | 30
VIIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0
Vascular encephalopathy (Nervous system disorders) | 1 | 0 | 0
Vertebral artery dissection (Nervous system disorders) | 0 | 1 | 1
Vertebral artery stenosis (Nervous system disorders) | 0 | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 3 | 0 | 0
Vocal cord paresis (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 4 | 1 | 1
Completed suicide (Psychiatric disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 3 | 0
Delirium (Psychiatric disorders) | 0 | 2 | 1
Depression (Psychiatric disorders) | 5 | 1 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1 | 1
Mental status changes (Psychiatric disorders) | 4 | 1 | 1
Rapid eye movements sleep abnormal (Psychiatric disorders) | 0 | 1 | 0
Substance abuse (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 32 | 26 | 19
Acute prerenal failure (Renal and urinary disorders) | 2 | 1 | 0
Albuminuria (Renal and urinary disorders) | 1 | 0 | 0
Anuria (Renal and urinary disorders) | 1 | 0 | 1
Bladder neck sclerosis (Renal and urinary disorders) | 1 | 0 | 0
Bladder outlet obstruction (Renal and urinary disorders) | 0 | 1 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 4 | 1 | 2
Calculus urinary (Renal and urinary disorders) | 2 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 3 | 2 | 4
Cystitis glandularis (Renal and urinary disorders) | 0 | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0 | 0
Diabetic nephropathy (Renal and urinary disorders) | 2 | 2 | 2
Dysuria (Renal and urinary disorders) | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 4 | 2 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 2 | 0
Hypertensive nephropathy (Renal and urinary disorders) | 0 | 1 | 0
Lower urinary tract symptoms (Renal and urinary disorders) | 0 | 1 | 0
Microalbuminuria (Renal and urinary disorders) | 0 | 0 | 1
Nephritis (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 3 | 3 | 7
Nephropathy (Renal and urinary disorders) | 1 | 1 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 1
Obstructive uropathy (Renal and urinary disorders) | 0 | 1 | 1
Oliguria (Renal and urinary disorders) | 1 | 0 | 0
Polyuria (Renal and urinary disorders) | 1 | 0 | 0
Renal artery arteriosclerosis (Renal and urinary disorders) | 1 | 0 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 10 | 2 | 4
Renal impairment (Renal and urinary disorders) | 2 | 2 | 4
Renal infarct (Renal and urinary disorders) | 0 | 2 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 2
Urethral stenosis (Renal and urinary disorders) | 2 | 4 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 2 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 0 | 0
Urinary retention (Renal and urinary disorders) | 3 | 4 | 5
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 6 | 8 | 10
Cystocele (Reproductive system and breast disorders) | 0 | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 | 1 | 0
Genital prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 1
Prostatic obstruction (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatism (Reproductive system and breast disorders) | 0 | 0 | 2
Prostatitis (Reproductive system and breast disorders) | 2 | 2 | 2
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 1
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 3
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 11 | 6 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 6 | 9
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 4
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 6
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 2
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 1
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 4
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Vocal cord thickening (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 3
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Diabetic bullosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 12 | 10 | 11
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Leukoplakia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pemphigus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin fibrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 10 | 6 | 11
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Physical assault (Social circumstances) | 0 | 1 | 0
Angioplasty (Surgical and medical procedures) | 1 | 1 | 1
Coronary angioplasty (Surgical and medical procedures) | 3 | 0 | 2
Coronary arterial stent insertion (Surgical and medical procedures) | 1 | 2 | 1
Coronary artery bypass (Surgical and medical procedures) | 4 | 3 | 4
Coronary revascularisation (Surgical and medical procedures) | 5 | 2 | 4
Fracture treatment (Surgical and medical procedures) | 1 | 0 | 0
Percutaneous coronary intervention (Surgical and medical procedures) | 0 | 2 | 3
Prophylaxis (Surgical and medical procedures) | 1 | 0 | 0
Stent placement (Surgical and medical procedures) | 0 | 2 | 1
Accelerated hypertension (Vascular disorders) | 0 | 1 | 1
Aneurysm (Vascular disorders) | 0 | 0 | 1
Angiopathy (Vascular disorders) | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 1 | 3 | 4
Aortic arteriosclerosis (Vascular disorders) | 1 | 0 | 1
Aortic dissection (Vascular disorders) | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 4 | 2 | 3
Arterial disorder (Vascular disorders) | 4 | 0 | 1
Arterial haemorrhage (Vascular disorders) | 0 | 1 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 1 | 0
Arterial stenosis (Vascular disorders) | 3 | 1 | 0
Arteriosclerosis (Vascular disorders) | 2 | 1 | 1
Arteriovenous fistula (Vascular disorders) | 1 | 0 | 1
Arteritis (Vascular disorders) | 0 | 0 | 3
Deep vein thrombosis (Vascular disorders) | 5 | 3 | 10
Diabetic microangiopathy (Vascular disorders) | 1 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 1
Embolism arterial (Vascular disorders) | 0 | 0 | 1
Extremity necrosis (Vascular disorders) | 5 | 4 | 8
Femoral artery embolism (Vascular disorders) | 0 | 0 | 1
Femoral artery occlusion (Vascular disorders) | 1 | 3 | 5
Haematoma (Vascular disorders) | 0 | 1 | 2
Haemorrhage (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 10 | 4 | 7
Hypertensive crisis (Vascular disorders) | 8 | 3 | 4
Hypertensive emergency (Vascular disorders) | 2 | 0 | 0
Hypotension (Vascular disorders) | 9 | 5 | 4
Hypovolaemic shock (Vascular disorders) | 2 | 1 | 0
Iliac artery occlusion (Vascular disorders) | 1 | 0 | 2
Infarction (Vascular disorders) | 1 | 0 | 2
Intermittent claudication (Vascular disorders) | 2 | 4 | 5
Ischaemia (Vascular disorders) | 2 | 1 | 2
Leriche syndrome (Vascular disorders) | 1 | 0 | 0
Malignant hypertension (Vascular disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 2 | 3 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 23 | 28 | 30
Peripheral artery aneurysm (Vascular disorders) | 1 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 6 | 3 | 9
Peripheral artery thrombosis (Vascular disorders) | 0 | 1 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 1
Peripheral embolism (Vascular disorders) | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 9 | 4 | 11
Peripheral vascular disorder (Vascular disorders) | 8 | 3 | 6
Peripheral venous disease (Vascular disorders) | 1 | 0 | 0
Subclavian artery stenosis (Vascular disorders) | 0 | 1 | 1
Thrombophlebitis (Vascular disorders) | 2 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 2 | 2 | 2
Varicose ulceration (Vascular disorders) | 1 | 0 | 1
Varicose vein (Vascular disorders) | 2 | 0 | 1
Vascular calcification (Vascular disorders) | 1 | 1 | 0
Vascular insufficiency (Vascular disorders) | 0 | 0 | 1
Venous occlusion (Vascular disorders) | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 1 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=2333) | Empagliflozin 10 mg (N=2345) | Empagliflozin 25 mg (N=2342)
Constipation (Gastrointestinal disorders) | 109 | 91 | 119
Diarrhoea (Gastrointestinal disorders) | 171 | 145 | 144
Oedema peripheral (General disorders) | 155 | 84 | 75
Bronchitis (Infections and infestations) | 164 | 129 | 117
Influenza (Infections and infestations) | 165 | 134 | 149
Nasopharyngitis (Infections and infestations) | 217 | 210 | 220
Upper respiratory tract infection (Infections and infestations) | 199 | 191 | 175
Urinary tract infection (Infections and infestations) | 344 | 339 | 337
Hyperglycaemia (Metabolism and nutrition disorders) | 423 | 217 | 202
Hypoglycaemia (Metabolism and nutrition disorders) | 685 | 694 | 673
Arthralgia (Musculoskeletal and connective tissue disorders) | 130 | 107 | 148
Back pain (Musculoskeletal and connective tissue disorders) | 148 | 149 | 166
Pain in extremity (Musculoskeletal and connective tissue disorders) | 133 | 114 | 101
Dizziness (Nervous system disorders) | 151 | 170 | 173
Headache (Nervous system disorders) | 123 | 100 | 124
Cough (Respiratory, thoracic and mediastinal disorders) | 146 | 119 | 108
Hypertension (Vascular disorders) | 210 | 154 | 176

LIMITATIONS AND CAVEATS:
2 sets of duplicates(4 patients(pts)) were counted only once.652 sites were initiated and 611 enrolled.One site transferred all pts to other sites.27 pts randomised and 13 pts screened were excluded from analyses due to serious non-compliance

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights